CLINICAL TRIAL: NCT01026038
Title: A Phase 3, Open-label Study to Evaluate Persistence of the Antibody Response Elicited by Pneumococcal Conjugate Vaccine in Healthy Children Who Have Been Previously Immunized With a 4-Dose Series of a Pneumococcal Conjugate Vaccine During Infancy in Study 6096A1-008-EU and the Safety and Immunogenicity of 13-valent Pneumococcal Conjugate Vaccine Administered at Least 24 Months After the Last Toddler Dose of Pneumococcal Conjugate Vaccine
Brief Title: Study Evaluating Antibody Response Of 13-Valent Pneumococcal Conjugate Vaccine (13vPnC) 24 Months After Toddler Dose.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 6096A1-3021; B1851016
Record Dates: First submitted 2009-12-02; First posted 2009-12-04 (Estimated); Results first posted 2012-02-08 (Estimated); Last update posted 2012-02-08 (Estimated); Status verified 2012-01

CONDITIONS: 13-valent Pneumococcal Vaccine; Immunization; Safety; Antibody Response
Keywords: Pneumococcal vaccine 13-valent

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): 1 dose (0.5 mL), IM of 13vPnC vaccine.
  Interventions: Biological: 13-valent pneumococcal conjugate vaccine

INTERVENTIONS:
Biological: 13-valent pneumococcal conjugate vaccine — All subjects will receive 1 dose (0.5 mL), IM of 13vPnC vaccine. (at least 24 months after toddler dose).

SUMMARY:
This is an open-label study (a study in which the doctors and participants know which drug or vaccine is being administered) in children who previously received a 4-dose series of a pneumococcal conjugate vaccine (PnC) during infancy in Study 6096A1-008-EU (NCT00366678). In this study, participants will receive an additional dose of 13-valent pneumococcal conjugate vaccine. The purpose of this study is to evaluate persistence, if any, of the antibody response by measuring any remaining pneumococcal antibodies since the previous study. This study will also evaluate the safety and immunogenicity of 13-valent pneumococcal conjugate vaccine when administered at least 24 months after the last dose of pneumococcal conjugate vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects at least 3 years of age, who received all 4 assigned doses of pneumococcal conjugate vaccine and completed Study 6096A1-008-EU (NCT00366678) for at least 24 months

Exclusion Criteria:

* Vaccination with any licensed or investigational pneumococcal vaccine since completion of Study 6096A1-008-EU(NCT00366678).
* History of culture-proven invasive disease caused by S pneumoniae since the completion of Study 6096A1-008-EU (NCT00366678).
* Previous anaphylactic reaction to any vaccine or vaccine-related component.
* Contraindication to vaccination

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2010-04; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (24):
- France (24):
  - Pfizer Investigational Site, Ancenis
  - Pfizer Investigational Site, Bondues
  - Pfizer Investigational Site, Brest
  - Pfizer Investigational Site, Châlons-en-Champagne
  - Pfizer Investigational Site, Draguignan
  - Pfizer Investigational Site, Essey-lès-Nancy
  - Pfizer Investigational Site, Écully
  - Pfizer Investigational Site, Floirac
  - Pfizer Investigational Site, Garges Les Gonesses
  - Pfizer Investigational Site, Joué-lès-Tours
  - Pfizer Investigational Site, Le Havre
  - Pfizer Investigational Site, Lingolsheim
  - Pfizer Investigational Site, Lyon
  - Pfizer Investigational Site, Maromme
  - Pfizer Investigational Site, Moûtiers
  - Pfizer Investigational Site, Nancy
  - Pfizer Investigational Site, Nice
  - Pfizer Investigational Site, Olonne-sur-Mer
  - Pfizer Investigational Site, Strasbourg
  - Pfizer Investigational Site, Talence
  - Pfizer Investigational Site, Thionville
  - Pfizer Investigational Site, Tours
  - Pfizer Investigational Site, Villers-lès-Nancy
  - Pfizer Investigational Site, Vitry-sur-Seine

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=6096A1-3021&StudyName=Study%20Evaluating%20Antibody%20Response%20Of%2013-Valent%20Pneumococcal%20Conjugate%20Vaccine%20%2813vPnC%29%2024%20months%20after%20toddler%20dose.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 263 participants who had received a 4-dose vaccination series of pneumococcal conjugate vaccine as part of study 6096A1-008 (NCT00366678) were enrolled for this study. Out of those 1 participant was a screen failure and was not included in results.
Groups:
- 13vPnC/13vPnC/13vPnC: Single dose (0.5 milliliter [mL]) of 13-valent pneumococcal conjugate (13vPnC) vaccine intramuscularly (IM), 2 years after receiving a full schedule (3 infant doses/1 toddler dose) of 13vPnC/13vPnC vaccine.
- 7vPnC/7vPnC/13vPnC: Single dose (0.5 mL) of 13vPnC vaccine IM, 2 years after receiving a full schedule (3 infant doses/1 toddler dose) of 7-valent pneumococcal conjugate (7vPnC)/7vPnC vaccine.
- 7vPnC/13vPnC/13vPnC: Single dose (0.5 mL) of 13vPnC vaccine IM, 2 years after receiving a full schedule (3 infant doses/1 toddler dose) of 7vPnC/13vPnC vaccine.
Period: Overall Study
Arm/Group | 13vPnC/13vPnC/13vPnC | 7vPnC/7vPnC/13vPnC | 7vPnC/13vPnC/13vPnC
Started | 130 | 65 | 67
Completed | 129 | 64 | 67
Not Completed | 1 | 1 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 13vPnC/13vPnC/13vPnC | 7vPnC/7vPnC/13vPnC | 7vPnC/13vPnC/13vPnC | Total
Number analyzed (Participants) | 130 | 65 | 67 | 262
Age Continuous [Mean (Standard Deviation); unit: Years] | 3.4 (0.25) | 3.4 (0.24) | 3.5 (0.25) | 3.4 (0.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 29 | 40 | 139
  Male | 60 | 36 | 27 | 123

OUTCOME MEASURES:

1. Primary Outcome: Serotype-specific Pneumococcal Immunoglobulin G (IgG) Geometric Mean Concentration (GMC) 1 Month After Single Dose of 13 Valent Pneumococcal Conjugate (13vPnC) Vaccine
Description: Antibody GMC as measured by microgram/millilitre (mcg/mL) for 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (Serotypes 1, 3, 5, 6A, 7F, and 19A) are presented. GMC (13vPnC) and corresponding 2-sided 95% confidence intervals (CI) were evaluated. Geometric means (GMs) were calculated using all participants with available data for the specified blood draw.
Time Frame: One month after vaccination
Population: Evaluable immunogenicity population: eligible participants, randomized, blood drawn within required timeframes, at least 1 valid and determinate assay result for proposed analysis, received no prohibited vaccines, no major protocol violations. N= number of participants with determinate IgG antibody concentration to serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | 13vPnC/13vPnC/13vPnC | 7vPnC/7vPnC/13vPnC | 7vPnC/13vPnC/13vPnC
Number analyzed (Participants) | 120 | 57 | 58
mcg/mL
  4 | 10.34 [8.94 to 11.97] | 12.79 [10.00 to 16.35] | 8.98 [6.98 to 11.56]
  6B | 31.62 [27.02 to 37.01] | 51.07 [38.65 to 67.49] | 35.38 [27.25 to 45.93]
  9V | 6.76 [5.90 to 7.73] | 6.50 [5.31 to 7.95] | 6.19 [5.04 to 7.61]
  14 | 21.55 [18.41 to 25.24] | 21.15 [16.89 to 26.48] | 20.73 [16.45 to 26.12]
  18C | 4.56 [3.93 to 5.29] | 6.12 [4.89 to 7.65] | 5.35 [4.27 to 6.71]
  19F | 16.59 [13.57 to 20.28] | 12.07 [9.35 to 15.59] | 15.09 [11.17 to 20.39]
  23F | 8.68 [7.50 to 10.03] | 10.87 [8.30 to 14.22] | 9.10 [7.34 to 11.28]
  1 | 10.72 [9.17 to 12.52] | 2.96 [2.45 to 3.59] | 20.69 [16.14 to 26.53]
  3 | 1.81 [1.46 to 2.23] | 1.60 [1.19 to 2.17] | 2.07 [1.66 to 2.59]
  5 | 10.00 [8.63 to 11.58] | 2.86 [2.37 to 3.46] | 19.20 [14.93 to 24.70]
  6A | 23.09 [19.50 to 27.33] | 14.38 [10.53 to 19.64] | 18.60 [13.87 to 24.93]
  7F | 8.23 [7.11 to 9.52] | 5.04 [4.16 to 6.11] | 8.02 [6.66 to 9.67]
  19A | 17.10 [14.54 to 20.11] | 8.58 [6.70 to 10.99] | 16.46 [13.42 to 20.19]
Statistical Analysis 1: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; Serotype 4: CI for the GMC ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/13vPnC/13vPnC - 7vPnC/7vPnC/13vPnC); Test type: Superiority or Other; GMC ratio = 0.81, 95% CI 2-sided [0.61 to 1.07]
Statistical Analysis 2: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 4: CI for the GMC ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/13vPnC/13vPnC - 7vPnC/13vPnC/13vPnC); Test type: Superiority or Other; GMC Ratio = 1.15, 95% CI 2-sided [0.87 to 1.52]
Statistical Analysis 3: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 4: CI for the GMC ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (7vPnC/7vPnC/13vPnC - 7vPnC/13vPnC/13vPnC); Test type: Superiority or Other; GMC Ratio = 1.42, 95% CI 2-sided [1.03 to 1.96]
Statistical Analysis 4: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; Serotype 6B: CI for the GMC ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/13vPnC/13vPnC - 7vPnC/7vPnC/13vPnC); Test type: Superiority or Other; GMC ratio = 0.62, 95% CI 2-sided [0.46 to 0.84]
Statistical Analysis 5: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 6B: CI for the GMC ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/13vPnC/13vPnC - 7vPnC/13vPnC/13vPnC); Test type: Superiority or Other; GMC ratio = 0.89, 95% CI 2-sided [0.66 to 1.20]
Statistical Analysis 6: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 6B: CI for the GMC ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (7vPnC/7vPnC/13vPnC - 7vPnC/13vPnC/13vPnC); Test type: Superiority or Other; GMC ratio = 1.44, 95% CI 2-sided [1.02 to 2.04]
Statistical Analysis 7: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; Serotype 9V: CI for the GMC ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/13vPnC/13vPnC - 7vPnC/7vPnC/13vPnC); Test type: Superiority or Other; GMC ratio = 1.04, 95% CI 2-sided [0.82 to 1.32]
Statistical Analysis 8: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 9V: CI for the GMC ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/13vPnC/13vPnC - 7vPnC/13vPnC/13vPnC); Test type: Superiority or Other; GMC ratio = 1.09, 95% CI 2-sided [0.86 to 1.39]
Statistical Analysis 9: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 9V: CI for the GMC ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (7vPnC/7vPnC/13vPnC - 7vPnC/13vPnC/13vPnC); Test type: Superiority or Other; GMC ratio = 1.05, 95% CI 2-sided [0.79 to 1.39]
Statistical Analysis 10: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; Serotype 14: CI for the GMC ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/13vPnC/13vPnC - 7vPnC/7vPnC/13vPnC); Test type: Superiority or Other; GMC ratio = 1.02, 95% CI 2-sided [0.77 to 1.34]
Statistical Analysis 11: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 14: CI for the GMC ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/13vPnC/13vPnC - 7vPnC/13vPnC/13vPnC); Test type: Superiority or Other; GMC ratio = 1.04, 95% CI 2-sided [0.79 to 1.37]
Statistical Analysis 12: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 14: CI for the GMC ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (7vPnC/7vPnC/13vPnC - 7vPnC/13vPnC/13vPnC); Test type: Superiority or Other; GMC ratio = 1.02, 95% CI 2-sided [0.74 to 1.40]
Statistical Analysis 13: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; Serotype 18C: CI for the GMC ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/13vPnC/13vPnC - 7vPnC/7vPnC/13vPnC); Test type: Superiority or Other; GMC ratio = 0.75, 95% CI 2-sided [0.57 to 0.97]
Statistical Analysis 14: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 18C: CI for the GMC ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/13vPnC/13vPnC - 7vPnC/13vPnC/13vPnC); Test type: Superiority or Other; GMC ratio = 0.85, 95% CI 2-sided [0.65 to 1.11]
Statistical Analysis 15: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 18C: CI for the GMC ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (7vPnC/7vPnC/13vPnC - 7vPnC/13vPnC/13vPnC); Test type: Superiority or Other; GMCratio = 1.14, 95% CI 2-sided [0.84 to 1.56]
Statistical Analysis 16: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; Serotype 19F: CI for the GMC ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/13vPnC/13vPnC - 7vPnC/7vPnC/13vPnC); Test type: Superiority or Other; GMC ratio = 1.37, 95% CI 2-sided [0.97 to 1.94]
Statistical Analysis 17: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 19F: CI for the GMC ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/13vPnC/13vPnC - 7vPnC/13vPnC/13vPnC); Test type: Superiority or Other; GMC ratio = 1.10, 95% CI 2-sided [0.78 to 1.55]
Statistical Analysis 18: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 19F: CI for the GMC ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (7vPnC/7vPnC/13vPnC - 7vPnC/13vPnC/13vPnC); Test type: Superiority or Other; GMC ratio = 0.80, 95% CI 2-sided [0.54 to 1.19]
Statistical Analysis 19: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; Serotype 23F: CI for the GMC ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/13vPnC/13vPnC - 7vPnC/7vPnC/13vPnC); Test type: Superiority or Other; GMC ratio = 0.80, 95% CI 2-sided [0.61 to 1.05]
Statistical Analysis 20: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 23F: CI for the GMC ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/13vPnC/13vPnC - 7vPnC/13vPnC/13vPnC); Test type: Superiority or Other; GMC ratio = 0.95, 95% CI 2-sided [0.73 to 1.25]
Statistical Analysis 21: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 23F: CI for the GMC ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (7vPnC/7vPnC/13vPnC - 7vPnC/13vPnC/13vPnC); Test type: Superiority or Other; GMC ratio = 1.19, 95% CI 2-sided [0.87 to 1.64]
Statistical Analysis 22: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; Serotype 1: CI for the GMC ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/13vPnC/13vPnC - 7vPnC/7vPnC/13vPnC); Test type: Superiority or Other; GMC ratio = 3.62, 95% CI 2-sided [2.76 to 4.74]
Statistical Analysis 23: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 1: CI for the GMC ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/13vPnC/13vPnC - 7vPnC/13vPnC/13vPnC); Test type: Superiority or Other; GMC ratio = 0.52, 95% CI 2-sided [0.40 to 0.68]
Statistical Analysis 24: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 1: CI for the GMC ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (7vPnC/7vPnC/13vPnC - 7vPnC/13vPnC/13vPnC); Test type: Superiority or Other; GMC ratio = 0.14, 95% CI 2-sided [0.10 to 0.20]
Statistical Analysis 25: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; Serotype 3: CI for the GMC ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/13vPnC/13vPnC - 7vPnC/7vPnC/13vPnC); Test type: Superiority or Other; GMC ratio = 1.13, 95% CI 2-sided [0.80 to 1.59]
Statistical Analysis 26: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 3: CI for the GMC ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/13vPnC/13vPnC - 7vPnC/13vPnC/13vPnC); Test type: Superiority or Other; GMC ratio = 0.87, 95% CI 2-sided [0.62 to 1.23]
Statistical Analysis 27: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 3: CI for the GMC ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (7vPnC/7vPnC/13vPnC - 7vPnC/13vPnC/13vPnC); Test type: Superiority or Other; GMC ratio = 0.77, 95% CI 2-sided [0.52 to 1.15]
Statistical Analysis 28: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; Serotype 5: CI for the GMC ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/13vPnC/13vPnC - 7vPnC/7vPnC/13vPnC); Test type: Superiority or Other; GMC ratio = 3.49, 95% CI 2-sided [2.68 to 4.54]
Statistical Analysis 29: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 5: CI for the GMC ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/13vPnC/13vPnC - 7vPnC/13vPnC/13vPnC); Test type: Superiority or Other; GMC ratio = 0.52, 95% CI 2-sided [0.40 to 0.68]
Statistical Analysis 30: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 5: CI for the GMC ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (7vPnC/7vPnC/13vPnC - 7vPnC/13vPnC/13vPnC); Test type: Superiority or Other; GMC ratio = 0.15, 95% CI 2-sided [0.11 to 0.20]
Statistical Analysis 31: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; Serotype 6A: CI for the GMC ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/13vPnC/13vPnC - 7vPnC/7vPnC/13vPnC); Test type: Superiority or Other; GMC ratio = 1.61, 95% CI 2-sided [1.15 to 2.23]
Statistical Analysis 32: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 6A: CI for the GMC ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/13vPnC/13vPnC - 7vPnC/13vPnC/13vPnC); Test type: Superiority or Other; GMC ratio = 1.24, 95% CI 2-sided [0.89 to 1.72]
Statistical Analysis 33: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 6A: CI for the GMC ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (7vPnC/7vPnC/13vPnC - 7vPnC/13vPnC/13vPnC); Test type: Superiority or Other; GMC ratio = 0.77, 95% CI 2-sided [0.53 to 1.13]
Statistical Analysis 34: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; Serotype 7F: CI for the GMC ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/13vPnC/13vPnC - 7vPnC/7vPnC/13vPnC); Test type: Superiority or Other; GMC ratio = 1.63, 95% CI 2-sided [1.28 to 2.08]
Statistical Analysis 35: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 7F: CI for the GMC ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/13vPnC/13vPnC - 7vPnC/13vPnC/13vPnC); Test type: Superiority or Other; GMC ratio = 1.03, 95% CI 2-sided [0.81 to 1.30]
Statistical Analysis 36: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 7F: CI for the GMC ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (7vPnC/7vPnC/13vPnC - 7vPnC/13vPnC/13vPnC); Test type: Superiority or Other; GMC ratio = 0.63, 95% CI 2-sided [0.47 to 0.83]
Statistical Analysis 37: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; Serotype 19A: CI for the GMC ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/13vPnC/13vPnC - 7vPnC/7vPnC/13vPnC); Test type: Superiority or Other; GMC ratio = 1.99, 95% CI 2-sided [1.51 to 2.63]
Statistical Analysis 38: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 19A: CI for the GMC ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/13vPnC/13vPnC - 7vPnC/13vPnC/13vPnC); Test type: Superiority or Other; GMC ratio = 1.04, 95% CI 2-sided [0.79 to 1.37]
Statistical Analysis 39: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 19A: CI for the GMC ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (7vPnC/7vPnC/13vPnC - 7vPnC/13vPnC/13vPnC); Test type: Superiority or Other; GMC ratio = 0.52, 95% CI 2-sided [0.38 to 0.72]

2. Primary Outcome: Percentage of Participants With Prespecified Local Reactions
Description: Local reactions (redness, swelling and pain) were reported using electronic diary. Redness and swelling were recorded in caliper units (range 1 to 14+), each caliper unit represented 0.5 cm. Categorized as any, absent (no redness or swelling present; 0 caliper units), mild (0.5 to 2.0 cm; 1 to 4 caliper units); moderate (2.5 to 7.0 cm; 5 to 14 caliper units); or severe (>7.0 cm; >14 caliper units). Pain was categorized as any, mild: does not interfere with activity; moderate: interferes with activity; severe: prevents daily activity. Participants may be reported in more than 1 category.
Time Frame: Seven days after vaccination
Population: Safety population: all participants who received the single dose of 13vPnC vaccination. "n" is signifying number of participants reporting yes for at least 1 day or no for all days, for each group, respectively.
Measure: Number; unit: Percentage of Participants
Arm/Group | 13vPnC/13vPnC/13vPnC | 7vPnC/7vPnC/13vPnC | 7vPnC/13vPnC/13vPnC
Number analyzed (Participants) | 130 | 64 | 64
Percentage of Participants
  Pain: Any (n= 112, 52, 53) | 55.4 | 55.8 | 64.2
  Pain: Mild (n= 109, 51, 51) | 50.5 | 49.0 | 56.9
  Pain: Moderate (n= 95, 47, 48) | 17.9 | 25.5 | 20.8
  Pain: Severe (n= 90, 43, 45) | 1.1 | 2.3 | 2.2
  Swelling: Any (101, 48, 47) | 39.6 | 41.7 | 27.7
  Swelling: Mild (n= 96, 48, 47) | 28.1 | 35.4 | 23.4
  Swelling: Moderate (n= 97, 44, 46) | 24.7 | 20.5 | 10.9
  Swelling: Severe (n= 90, 43, 45) | 0.0 | 2.3 | 0.0
  Redness: Any (n= 105, 50, 50) | 48.6 | 54.0 | 46.0
  Redness: Mild (n= 101, 49, 48) | 38.6 | 40.8 | 37.5
  Redness: Moderate (n= 95, 45, 47) | 22.1 | 31.1 | 17.0
  Redness: Severe (n= 90, 43, 45) | 0.0 | 2.3 | 0.0
Statistical Analysis 1: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; Pain (Any): Fisher exact test, 2-sided was used. Pairwise comparison was made between 13vPnC/13vPnC/13vPnC and 7vPnC/7vPnC/13vPnC; Test type: Superiority or Other; p > 0.990, Fisher Exact
Statistical Analysis 2: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Pain (Any): Fisher exact test, 2-sided was used. Pairwise comparison was made between 7vPnC/7vPnC/13vPnC and 7vPnC/13vPnC/13vPnC; Test type: Superiority or Other; p = 0.429, Fisher Exact
Statistical Analysis 3: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Pain (Any): Fisher exact test, 2-sided was used. Pairwise comparison was made between 13vPnC/13vPnC/13vPnC and 7vPnC/13vPnC/13vPnC; Test type: Superiority or Other; p = 0.314, Fisher Exact
Statistical Analysis 4: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; Pain (Mild): Fisher exact test, 2-sided was used. Pairwise comparison was made between 13vPnC/13vPnC/13vPnC and 7vPnC/7vPnC/13vPnC; Test type: Superiority or Other; p > 0.990, Fisher Exact
Statistical Analysis 5: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Pain (Mild): Fisher exact test, 2-sided was used. Pairwise comparison was made between 7vPnC/7vPnC/13vPnC and 7vPnC/13vPnC/13vPnC; Test type: Superiority or Other; p = 0.552, Fisher Exact
Statistical Analysis 6: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Pain (Mild): Fisher exact test, 2-sided was used. Pairwise comparison was made between 13vPnC/13vPnC/13vPnC and 7vPnC/13vPnC/13vPnC; Test type: Superiority or Other; p = 0.499, Fisher Exact
Statistical Analysis 7: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; Pain (Moderate): Fisher exact test, 2-sided was used. Pairwise comparison was made between 13vPnC/13vPnC/13vPnC and 7vPnC/7vPnC/13vPnC; Test type: Superiority or Other; p = 0.376, Fisher Exact
Statistical Analysis 8: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Pain (Moderate): Fisher exact test, 2-sided was used. Pairwise comparison was made between 7vPnC/7vPnC/13vPnC and 7vPnC/13vPnC/13vPnC; Test type: Superiority or Other; p = 0.633, Fisher Exact
Statistical Analysis 9: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Pain (Moderate): Fisher exact test, 2-sided was used. Pairwise comparison was made between 13vPnC/13vPnC/13vPnC and 7vPnC/13vPnC/13vPnC; Test type: Superiority or Other; p = 0.658, Fisher Exact
Statistical Analysis 10: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; Pain (Severe): Fisher exact test, 2-sided was used. Pairwise comparison was made between 13vPnC/13vPnC/13vPnC and 7vPnC/7vPnC/13vPnC; Test type: Superiority or Other; p = 0.544, Fisher Exact
Statistical Analysis 11: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Pain (Severe): Fisher exact test, 2-sided was used. Pairwise comparison was made between 7vPnC/7vPnC/13vPnC and 7vPnC/13vPnC/13vPnC; Test type: Superiority or Other; p > 0.990, Fisher Exact
Statistical Analysis 12: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Pain (Severe): Fisher exact test, 2-sided was used. Pairwise comparison was made between 13vPnC/13vPnC/13vPnC and 7vPnC/13vPnC/13vPnC; Test type: Superiority or Other; p > 0.990, Fisher Exact
Statistical Analysis 13: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; Swelling (Any): Fisher exact test, 2-sided was used. Pairwise comparison was made between 13vPnC/13vPnC/13vPnC and 7vPnC/7vPnC/13vPnC; Test type: Superiority or Other; p = 0.859, Fisher Exact
Statistical Analysis 14: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Swelling (Any): Fisher exact test, 2-sided was used. Pairwise comparison was made between 7vPnC/7vPnC/13vPnC and 7vPnC/13vPnC/13vPnC; Test type: Superiority or Other; p = 0.197, Fisher Exact
Statistical Analysis 15: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Swelling (Any): Fisher exact test, 2-sided was used. Pairwise comparison was made between 13vPnC/13vPnC/13vPnC and 7vPnC/13vPnC/13vPnC; Test type: Superiority or Other; p = 0.198, Fisher Exact
Statistical Analysis 16: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; Swelling (Mild): Fisher exact test, 2-sided was used. Pairwise comparison was made between 13vPnC/13vPnC/13vPnC and 7vPnC/7vPnC/13vPnC; Test type: Superiority or Other; p = 0.443, Fisher Exact
Statistical Analysis 17: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Swelling (Mild): Fisher exact test, 2-sided was used. Pairwise comparison was made between 7vPnC/7vPnC/13vPnC and 7vPnC/13vPnC/13vPnC; Test type: Superiority or Other; p = 0.261, Fisher Exact
Statistical Analysis 18: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Swelling (Mild): Fisher exact test, 2-sided was used. Pairwise comparison was made between 13vPnC/13vPnC/13vPnC and 7vPnC/13vPnC/13vPnC; Test type: Superiority or Other; p = 0.687, Fisher Exact
Statistical Analysis 19: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; Swelling (Moderate): Fisher exact test, 2-sided was used. Pairwise comparison was made between 13vPnC/13vPnC/13vPnC and 7vPnC/7vPnC/13vPnC; Test type: Superiority or Other; p = 0.671, Fisher Exact
Statistical Analysis 20: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Swelling (Moderate): Fisher exact test, 2-sided was used. Pairwise comparison was made between 7vPnC/7vPnC/13vPnC and 7vPnC/13vPnC/13vPnC; Test type: Superiority or Other; p = 0.253, Fisher Exact
Statistical Analysis 21: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Swelling (Moderate): Fisher exact test, 2-sided was used. Pairwise comparison was made between 13vPnC/13vPnC/13vPnC and 7vPnC/13vPnC/13vPnC; Test type: Superiority or Other; p = 0.074, Fisher Exact
Statistical Analysis 22: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; Swelling (Severe): Fisher exact test, 2-sided was used. Pairwise comparison was made between 13vPnC/13vPnC/13vPnC and 7vPnC/7vPnC/13vPnC; Test type: Superiority or Other; p = 0.323, Fisher Exact
Statistical Analysis 23: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Swelling (Severe): Fisher exact test, 2-sided was used. Pairwise comparison was made between 7vPnC/7vPnC/13vPnC and 7vPnC/13vPnC/13vPnC; Test type: Superiority or Other; p = 0.489, Fisher Exact
Statistical Analysis 24: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; Redness (Any): Fisher exact test, 2-sided was used. Pairwise comparison was made between 13vPnC/13vPnC/13vPnC and 7vPnC/7vPnC/13vPnC; Test type: Superiority or Other; p = 0.607, Fisher Exact
Statistical Analysis 25: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Redness (Any): Fisher exact test, 2-sided was used. Pairwise comparison was made between 7vPnC/7vPnC/13vPnC and 7vPnC/13vPnC/13vPnC; Test type: Superiority or Other; p = 0.549, Fisher Exact
Statistical Analysis 26: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Redness (Any): Fisher exact test, 2-sided was used. Pairwise comparison was made between 13vPnC/13vPnC/13vPnC and 7vPnC/13vPnC/13vPnC; Test type: Superiority or Other; p = 0.864, Fisher Exact
Statistical Analysis 27: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; Redness (Mild): Fisher exact test, 2-sided was used. Pairwise comparison was made between 13vPnC/13vPnC/13vPnC and 7vPnC/7vPnC/13vPnC; Test type: Superiority or Other; p = 0.859, Fisher Exact
Statistical Analysis 28: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Redness (Mild): Fisher exact test, 2-sided was used. Pairwise comparison was made between 7vPnC/7vPnC/13vPnC and 7vPnC/13vPnC/13vPnC; Test type: Superiority or Other; p = 0.836, Fisher Exact
Statistical Analysis 29: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Redness (Mild): Fisher exact test, 2-sided was used. Pairwise comparison was made between 13vPnC/13vPnC/13vPnC and 7vPnC/13vPnC/13vPnC; Test type: Superiority or Other; p > 0.990, Fisher Exact
Statistical Analysis 30: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; Redness (Moderate): Fisher exact test, 2-sided was used. Pairwise comparison was made between 13vPnC/13vPnC/13vPnC and 7vPnC/7vPnC/13vPnC; Test type: Superiority or Other; p = 0.297, Fisher Exact
Statistical Analysis 31: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Redness (Moderate): Fisher exact test, 2-sided was used. Pairwise comparison was made between 7vPnC/7vPnC/13vPnC and 7vPnC/13vPnC/13vPnC; Test type: Superiority or Other; p = 0.145, Fisher Exact
Statistical Analysis 32: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Redness (Moderate): Fisher exact test, 2-sided was used. Pairwise comparison was made between 13vPnC/13vPnC/13vPnC and 7vPnC/13vPnC/13vPnC; Test type: Superiority or Other; p = 0.517, Fisher Exact
Statistical Analysis 33: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; Redness (Severe): Fisher exact test, 2-sided was used. Pairwise comparison was made between 13vPnC/13vPnC/13vPnC and 7vPnC/7vPnC/13vPnC; Test type: Superiority or Other; p = 0.323, Fisher Exact
Statistical Analysis 34: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Redness (Severe): Fisher exact test, 2-sided was used. Pairwise comparison was made between 7vPnC/7vPnC/13vPnC and 7vPnC/13vPnC/13vPnC; Test type: Superiority or Other; p = 0.489, Fisher Exact

3. Primary Outcome: Percentage of Participants With Prespecified Systemic Events
Description: Systemic events (any fever >= 38 degree celsius [C], vomiting, diarrhea, and fatigue) were reported using electronic diary. Fever categorized as >=38 to <=39 degree C; >39 to <=40 degree C; >40 degree C. Vomiting: mild (1-2 times/day ); moderate (>2 times/day); severe (requires intravenous hydration). Diarrhea: mild (2-3 loose stools/day); moderate (4-5 stools/day); severe (>=6 loose stools/day). Fatigue: mild (does not interfere with activity); moderate (some interference with activity); severe (prevents daily routine activity). Participants may be reported in more than 1 category.
Time Frame: Seven days after vaccination
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | 13vPnC/13vPnC/13vPnC | 7vPnC/7vPnC/13vPnC | 7vPnC/13vPnC/13vPnC
Number analyzed (Participants) | 130 | 64 | 64
Percentage of Participants
  Fever >=38 to <=39 degree C (n= 93, 49, 46) | 15.1 | 28.6 | 19.6
  Fever >39 to <=40 degree C (n= 92, 43, 46) | 2.2 | 4.7 | 2.2
  Fever >40 degree C (n= 90, 43, 45) | 0.0 | 0.0 | 2.2
  Vomiting: Any (n= 91, 44, 45) | 3.3 | 9.1 | 6.7
  Vomiting: Mild (n= 91, 44, 45) | 3.3 | 9.1 | 6.7
  Vomiting: Moderate (n= 90, 43, 45) | 0.0 | 0.0 | 0.0
  Vomiting: Severe (n= 90, 43, 45) | 0.0 | 0.0 | 0.0
  Diarrhea: Any (n= 90, 45, 47) | 8.9 | 17.8 | 8.5
  Diarrhea: Mild (n= 90, 45, 47) | 8.9 | 17.8 | 8.5
  Diarrhea: Moderate (n= 90, 43, 45) | 1.1 | 0.0 | 0.0
  Diarrhea: Severe (n= 90, 43, 45) | 0.0 | 0.0 | 0.0
  Fatigue: Any (n= 103, 54, 48) | 40.8 | 51.9 | 31.3
  Fatigue: Mild (n= 100, 49, 48) | 34.0 | 34.7 | 20.8
  Fatigue: Moderate (n= 96, 49, 46) | 16.7 | 30.6 | 15.2
  Fatigue: Severe (n= 92, 43, 45) | 3.3 | 2.3 | 2.2
Statistical Analysis 1: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; Fever (>=38 degree C to <=39 degree C): Fisher exact test, 2-sided was used. Pairwise comparison was made between 13vPnC/13vPnC/13vPnC and 7vPnC/7vPnC/13vPnC; Test type: Superiority or Other; p = 0.075, Fisher Exact
Statistical Analysis 2: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Fever (>=38 degree C to <=39 degree C): Fisher exact test, 2-sided was used. Pairwise comparison was made between 7vPnC/7vPnC/13vPnC and 7vPnC/13vPnC/13vPnC; Test type: Superiority or Other; p = 0.345, Fisher Exact
Statistical Analysis 3: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Fever (>=38 degree C to <=39 degree C): Fisher exact test, 2-sided was used. Pairwise comparison was made between 13vPnC/13vPnC/13vPnC and 7vPnC/13vPnC/13vPnC; Test type: Superiority or Other; p = 0.628, Fisher Exact
Statistical Analysis 4: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; Fever (>=39 degree C to <=40 degree C): Fisher exact test, 2-sided was used. Pairwise comparison was made between 13vPnC/13vPnC/13vPnC and 7vPnC/7vPnC/13vPnC; Test type: Superiority or Other; p = 0.592, Fisher Exact
Statistical Analysis 5: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Fever (>=39 degree C to <=40 degree C): Fisher exact test, 2-sided was used. Pairwise comparison was made between 7vPnC/7vPnC/13vPnC and 7vPnC/13vPnC/13vPnC; Test type: Superiority or Other; p = 0.608, Fisher Exact
Statistical Analysis 6: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Fever (>=39 degree C to <=40 degree C): Fisher exact test, 2-sided was used. Pairwise comparison was made between 13vPnC/13vPnC/13vPnC and 7vPnC/13vPnC/13vPnC; Test type: Superiority or Other; p > 0.990, Fisher Exact
Statistical Analysis 7: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Fever (>40 degree C): Fisher exact test, 2-sided was used. Pairwise comparison was made between 7vPnC/7vPnC/13vPnC and 7vPnC/13vPnC/13vPnC; Test type: Superiority or Other; p > 0.990, Fisher Exact
Statistical Analysis 8: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Fever (>40 degree C): Fisher exact test, 2-sided was used. Pairwise comparison was made between 13vPnC/13vPnC/13vPnC and 7vPnC/13vPnC/13vPnC; Test type: Superiority or Other; p = 0.333, Fisher Exact
Statistical Analysis 9: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; Vomiting (Any): Fisher exact test, 2-sided was used. Pairwise comparison was made between 13vPnC/13vPnC/13vPnC and 7vPnC/7vPnC/13vPnC; Test type: Superiority or Other; p = 0.215, Fisher Exact
Statistical Analysis 10: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Vomiting (Any): Fisher exact test, 2-sided was used. Pairwise comparison was made between 7vPnC/7vPnC/13vPnC and 7vPnC/13vPnC/13vPnC; Test type: Superiority or Other; p = 0.714, Fisher Exact
Statistical Analysis 11: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Vomiting (Any): Fisher exact test, 2-sided was used. Pairwise comparison was made between 13vPnC/13vPnC/13vPnC and 7vPnC/13vPnC/13vPnC; Test type: Superiority or Other; p = 0.397, Fisher Exact
Statistical Analysis 12: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; Vomiting (Mild): Fisher exact test, 2-sided was used. Pairwise comparison was made between 13vPnC/13vPnC/13vPnC and 7vPnC/7vPnC/13vPnC; Test type: Superiority or Other; p = 0.215, Fisher Exact
Statistical Analysis 13: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Vomiting (Mild): Fisher exact test, 2-sided was used. Pairwise comparison was made between 7vPnC/7vPnC/13vPnC and 7vPnC/13vPnC/13vPnC; Test type: Superiority or Other; p = 0.714, Fisher Exact
Statistical Analysis 14: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Vomiting (Mild): Fisher exact test, 2-sided was used. Pairwise comparison was made between 13vPnC/13vPnC/13vPnC and 7vPnC/13vPnC/13vPnC; Test type: Superiority or Other; p = 0.397, Fisher Exact
Statistical Analysis 15: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; Diarrhea (Any): Fisher exact test, 2-sided was used. Pairwise comparison was made between 13vPnC/13vPnC/13vPnC and 7vPnC/7vPnC/13vPnC; Test type: Superiority or Other; p = 0.161, Fisher Exact
Statistical Analysis 16: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Diarrhea (Any): Fisher exact test, 2-sided was used. Pairwise comparison was made between 7vPnC/7vPnC/13vPnC and 7vPnC/13vPnC/13vPnC; Test type: Superiority or Other; p = 0.226, Fisher Exact
Statistical Analysis 17: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Diarrhea (Any): Fisher exact test, 2-sided was used. Pairwise comparison was made between 13vPnC/13vPnC/13vPnC and 7vPnC/13vPnC/13vPnC; Test type: Superiority or Other; p > 0.990, Fisher Exact
Statistical Analysis 18: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; Diarrhea (Mild): Fisher exact test, 2-sided was used. Pairwise comparison was made between 13vPnC/13vPnC/13vPnC and 7vPnC/7vPnC/13vPnC; Test type: Superiority or Other; p = 0.161, Fisher Exact
Statistical Analysis 19: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Diarrhea (Mild): Fisher exact test, 2-sided was used. Pairwise comparison was made between 7vPnC/7vPnC/13vPnC and 7vPnC/13vPnC/13vPnC; Test type: Superiority or Other; p = 0.226, Fisher Exact
Statistical Analysis 20: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Diarrhea (Mild): Fisher exact test, 2-sided was used. Pairwise comparison was made between 13vPnC/13vPnC/13vPnC and 7vPnC/13vPnC/13vPnC; Test type: Superiority or Other; p > 0.990, Fisher Exact
Statistical Analysis 21: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; Diarrhea (Moderate): Fisher exact test, 2-sided was used. Pairwise comparison was made between 13vPnC/13vPnC/13vPnC and 7vPnC/7vPnC/13vPnC; Test type: Superiority or Other; p > 0.990, Fisher Exact
Statistical Analysis 22: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Diarrhea (Moderate): Fisher exact test, 2-sided was used. Pairwise comparison was made between 13vPnC/13vPnC/13vPnC and 7vPnC/13vPnC/13vPnC; Test type: Superiority or Other; p > 0.990, Fisher Exact
Statistical Analysis 23: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; Fatigue (Any): Fisher exact test, 2-sided was used. Pairwise comparison was made between 13vPnC/13vPnC/13vPnC and 7vPnC/7vPnC/13vPnC; Test type: Superiority or Other; p = 0.237, Fisher Exact
Statistical Analysis 24: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Fatigue (Any): Fisher exact test, 2-sided was used. Pairwise comparison was made between 7vPnC/7vPnC/13vPnC and 7vPnC/13vPnC/13vPnC; Test type: Superiority or Other; p = 0.045, Fisher Exact
Statistical Analysis 25: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Fatigue (Any): Fisher exact test, 2-sided was used. Pairwise comparison was made between 13vPnC/13vPnC/13vPnC and 7vPnC/13vPnC/13vPnC; Test type: Superiority or Other; p = 0.285, Fisher Exact
Statistical Analysis 26: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; Fatigue (Mild): Fisher exact test, 2-sided was used. Pairwise comparison was made between 13vPnC/13vPnC/13vPnC and 7vPnC/7vPnC/13vPnC; Test type: Superiority or Other; p > 0.990, Fisher Exact
Statistical Analysis 27: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Fatigue (Mild): Fisher exact test, 2-sided was used. Pairwise comparison was made between 7vPnC/7vPnC/13vPnC and 7vPnC/13vPnC/13vPnC; Test type: Superiority or Other; p = 0.174, Fisher Exact
Statistical Analysis 28: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Fatigue (Mild): Fisher exact test, 2-sided was used. Pairwise comparison was made between 13vPnC/13vPnC/13vPnC and 7vPnC/13vPnC/13vPnC; Test type: Superiority or Other; p = 0.125, Fisher Exact
Statistical Analysis 29: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; Fatigue (Moderate): Fisher exact test, 2-sided was used. Pairwise comparison was made between 13vPnC/13vPnC/13vPnC and 7vPnC/7vPnC/13vPnC; Test type: Superiority or Other; p = 0.058, Fisher Exact
Statistical Analysis 30: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Fatigue (Moderate): Fisher exact test, 2-sided was used. Pairwise comparison was made between 7vPnC/7vPnC/13vPnC and 7vPnC/13vPnC/13vPnC; Test type: Superiority or Other; p = 0.092, Fisher Exact
Statistical Analysis 31: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Fatigue (Moderate): Fisher exact test, 2-sided was used. Pairwise comparison was made between 13vPnC/13vPnC/13vPnC and 7vPnC/13vPnC/13vPnC; Test type: Superiority or Other; p > 0.990, Fisher Exact
Statistical Analysis 32: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; Fatigue (Severe): Fisher exact test, 2-sided was used. Pairwise comparison was made between 13vPnC/13vPnC/13vPnC and 7vPnC/7vPnC/13vPnC; Test type: Superiority or Other; p > 0.990, Fisher Exact
Statistical Analysis 33: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Fatigue (Severe): Fisher exact test, 2-sided was used. Pairwise comparison was made between 7vPnC/7vPnC/13vPnC and 7vPnC/13vPnC/13vPnC; Test type: Superiority or Other; p > 0.990, Fisher Exact
Statistical Analysis 34: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Fatigue (Severe): Fisher exact test, 2-sided was used. Pairwise comparison was made between 13vPnC/13vPnC/13vPnC and 7vPnC/13vPnC/13vPnC; Test type: Superiority or Other; p > 0.990, Fisher Exact

4. Secondary Outcome: Serotype-specific Pneumococcal IgG GMC Prior to Single Dose of 13vPnC Vaccine
Description: IgG GMC to the 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) were determined in the blood samples of all the participants using a standardized anti-pneumococcal IgG enzymelinked immunosorbent assay (ELISA). CIs for GMC are back transformations of a CI based on the Student t distribution for the mean logarithm of the concentrations.
Time Frame: Up to 7 days before vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | 13vPnC/13vPnC/13vPnC | 7vPnC/7vPnC/13vPnC | 7vPnC/13vPnC/13vPnC
Number analyzed (Participants) | 120 | 57 | 58
mcg/mL
  4 | 0.17 [0.15 to 0.21] | 0.23 [0.18 to 0.30] | 0.18 [0.15 to 0.22]
  6B | 2.86 [2.35 to 3.48] | 4.10 [2.96 to 5.68] | 3.21 [2.37 to 4.36]
  9V | 0.72 [0.60 to 0.85] | 0.92 [0.72 to 1.17] | 0.71 [0.58 to 0.87]
  14 | 0.77 [0.61 to 0.98] | 0.74 [0.52 to 1.06] | 0.59 [0.42 to 0.83]
  18C | 0.21 [0.17 to 0.25] | 0.36 [0.28 to 0.47] | 0.23 [0.18 to 0.28]
  19F | 2.22 [1.67 to 2.95] | 2.11 [1.43 to 3.11] | 1.44 [1.04 to 2.02]
  23F | 1.26 [1.00 to 1.58] | 1.56 [1.19 to 2.05] | 1.18 [0.92 to 1.52]
  1 | 0.35 [0.29 to 0.43] | 0.14 [0.09 to 0.20] | 0.28 [0.23 to 0.34]
  3 | 0.50 [0.35 to 0.71] | 0.47 [0.29 to 0.75] | 0.42 [0.30 to 0.58]
  5 | 1.28 [1.07 to 1.53] | 1.12 [0.89 to 1.41] | 1.41 [1.19 to 1.67]
  6A | 4.05 [3.25 to 5.04] | 1.89 [1.50 to 2.38] | 2.47 [1.91 to 3.21]
  7F | 0.65 [0.55 to 0.78] | 0.21 [0.15 to 0.30] | 0.77 [0.62 to 0.96]
  19A | 6.16 [4.88 to 7.79] | 3.38 [2.60 to 4.41] | 4.63 [3.43 to 6.26]
Statistical Analysis 1: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; GMC ratio = 0.75, 95% CI 2-sided [0.56 to 1.00]
Statistical Analysis 2: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; GMC Ratio = 0.96, 95% CI 2-sided [0.73 to 1.28]
Statistical Analysis 3: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; GMC Ratio = 1.29, 95% CI 2-sided [0.92 to 1.79]
Statistical Analysis 4: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; [analysis description as in outcome 1, analysis 4]; Test type: Superiority or Other; GMC ratio = 0.70, 95% CI 2-sided [0.49 to 1.00]
Statistical Analysis 5: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 1, analysis 5]; Test type: Superiority or Other; GMC ratio = 0.89, 95% CI 2-sided [0.62 to 1.27]
Statistical Analysis 6: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 1, analysis 6]; Test type: Superiority or Other; GMC ratio = 1.27, 95% CI 2-sided [0.84 to 1.94]
Statistical Analysis 7: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; [analysis description as in outcome 1, analysis 7]; Test type: Superiority or Other; GMC ratio = 0.78, 95% CI 2-sided [0.58 to 1.03]
Statistical Analysis 8: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 1, analysis 8]; Test type: Superiority or Other; GMC ratio = 1.01, 95% CI 2-sided [0.76 to 1.33]
Statistical Analysis 9: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 1, analysis 9]; Test type: Superiority or Other; GMC ratio = 1.29, 95% CI 2-sided [0.93 to 1.80]
Statistical Analysis 10: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; [analysis description as in outcome 1, analysis 10]; Test type: Superiority or Other; GMC ratio = 1.04, 95% CI 2-sided [0.69 to 1.58]
Statistical Analysis 11: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 1, analysis 11]; Test type: Superiority or Other; GMC ratio = 1.30, 95% CI 2-sided [0.86 to 1.97]
Statistical Analysis 12: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 1, analysis 12]; Test type: Superiority or Other; GMC ratio = 1.25, 95% CI 2-sided [0.77 to 2.03]
Statistical Analysis 13: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; [analysis description as in outcome 1, analysis 13]; Test type: Superiority or Other; GMC ratio = 0.58, 95% CI 2-sided [0.42 to 0.78]
Statistical Analysis 14: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 1, analysis 14]; Test type: Superiority or Other; GMC ratio = 0.91, 95% CI 2-sided [0.67 to 1.23]
Statistical Analysis 15: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 1, analysis 15]; Test type: Superiority or Other; GMC ratio = 1.58, 95% CI 2-sided [1.11 to 2.25]
Statistical Analysis 16: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; [analysis description as in outcome 1, analysis 16]; Test type: Superiority or Other; GMC ratio = 1.05, 95% CI 2-sided [0.66 to 1.68]
Statistical Analysis 17: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 1, analysis 17]; Test type: Superiority or Other; GMC ratio = 1.54, 95% CI 2-sided [0.97 to 2.44]
Statistical Analysis 18: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 1, analysis 18]; Test type: Superiority or Other; GMC ratio = 1.46, 95% CI 2-sided [0.85 to 2.51]
Statistical Analysis 19: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; [analysis description as in outcome 1, analysis 19]; Test type: Superiority or Other; GMC ratio = 0.80, 95% CI 2-sided [0.56 to 1.15]
Statistical Analysis 20: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 1, analysis 20]; Test type: Superiority or Other; GMC ratio = 1.06, 95% CI 2-sided [0.74 to 1.52]
Statistical Analysis 21: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 1, analysis 21]; Test type: Superiority or Other; GMC ratio = 1.32, 95% CI 2-sided [0.87 to 2.01]
Statistical Analysis 22: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; [analysis description as in outcome 1, analysis 22]; Test type: Superiority or Other; GMC ratio = 2.59, 95% CI 2-sided [1.80 to 3.73]
Statistical Analysis 23: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 1, analysis 23]; Test type: Superiority or Other; GMC ratio = 1.26, 95% CI 2-sided [0.88 to 1.79]
Statistical Analysis 24: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 1, analysis 24]; Test type: Superiority or Other; GMC ratio = 0.49, 95% CI 2-sided [0.32 to 0.74]
Statistical Analysis 25: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; [analysis description as in outcome 1, analysis 25]; Test type: Superiority or Other; GMC ratio = 1.06, 95% CI 2-sided [0.61 to 1.87]
Statistical Analysis 26: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 1, analysis 26]; Test type: Superiority or Other; GMC ratio = 1.19, 95% CI 2-sided [0.68 to 2.09]
Statistical Analysis 27: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 1, analysis 27]; Test type: Superiority or Other; GMC ratio = 1.12, 95% CI 2-sided [0.59 to 2.15]
Statistical Analysis 28: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; [analysis description as in outcome 1, analysis 28]; Test type: Superiority or Other; GMC ratio = 1.15, 95% CI 2-sided [0.87 to 1.52]
Statistical Analysis 29: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 1, analysis 29]; Test type: Superiority or Other; GMC ratio = 0.91, 95% CI 2-sided [0.69 to 1.20]
Statistical Analysis 30: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 1, analysis 30]; Test type: Superiority or Other; GMC ratio = 0.79, 95% CI 2-sided [0.57 to 1.10]
Statistical Analysis 31: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; [analysis description as in outcome 1, analysis 31]; Test type: Superiority or Other; GMC ratio = 2.14, 95% CI 2-sided [1.52 to 3.02]
Statistical Analysis 32: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 1, analysis 32]; Test type: Superiority or Other; GMC ratio = 1.64, 95% CI 2-sided [1.16 to 2.30]
Statistical Analysis 33: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 1, analysis 33]; Test type: Superiority or Other; GMC ratio = 0.76, 95% CI 2-sided [0.51 to 1.14]
Statistical Analysis 34: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; [analysis description as in outcome 1, analysis 34]; Test type: Superiority or Other; GMC ratio = 3.11, 95% CI 2-sided [2.23 to 4.33]
Statistical Analysis 35: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 1, analysis 35]; Test type: Superiority or Other; GMC ratio = 0.84, 95% CI 2-sided [0.61 to 1.17]
Statistical Analysis 36: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 1, analysis 36]; Test type: Superiority or Other; GMC ratio = 0.27, 95% CI 2-sided [0.19 to 0.40]
Statistical Analysis 37: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; [analysis description as in outcome 1, analysis 37]; Test type: Superiority or Other; GMC ratrio = 1.82, 95% CI 2-sided [1.25 to 2.66]
Statistical Analysis 38: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 1, analysis 38]; Test type: Superiority or Other; GMC ratio = 1.33, 95% CI 2-sided [0.91 to 1.94]
Statistical Analysis 39: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 1, analysis 39]; Test type: Superiority or Other; GMC ratio = 0.73, 95% CI 2-sided [0.47 to 1.13]

5. Secondary Outcome: Serotype-specific Pneumococcal IgG GMC at 4 to 7 Days After the Single Dose of 13vPnC Vaccine
Description: IgG GMC to the 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) were determined in the blood samples of all the participants using a standardized anti-pneumococcal IgG ELISA. CIs for GMC are back transformations of a CI based on the Student t distribution for the mean logarithm of the concentrations.
Time Frame: Four to seven days after vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | 13vPnC/13vPnC/13vPnC | 7vPnC/7vPnC/13vPnC | 7vPnC/13vPnC/13vPnC
Number analyzed (Participants) | 44 | 18 | 22
mcg/mL
  4 | 2.96 [1.67 to 5.24] | 4.66 [2.01 to 10.82] | 3.85 [1.70 to 8.74]
  6B | 17.78 [12.50 to 25.30] | 19.15 [8.84 to 41.48] | 16.26 [8.10 to 32.66]
  9V | 3.49 [2.39 to 5.09] | 3.15 [1.75 to 5.66] | 3.20 [1.86 to 5.50]
  14 | 5.55 [3.32 to 9.30] | 5.67 [2.29 to 13.99] | 4.52 [2.14 to 9.52]
  18C | 2.31 [1.36 to 3.91] | 3.34 [1.66 to 6.72] | 2.51 [1.33 to 4.73]
  19F | 11.70 [7.21 to 19.00] | 6.88 [2.98 to 15.86] | 8.51 [4.38 to 16.55]
  23F | 5.24 [3.49 to 7.87] | 5.82 [2.97 to 11.40] | 6.28 [3.50 to 11.26]
  1 | 4.24 [2.48 to 7.26] | 0.56 [0.27 to 1.18] | 8.00 [3.51 to 18.23]
  3 | 1.24 [0.79 to 1.95] | 1.12 [0.56 to 2.25] | 1.24 [0.90 to 1.72]
  5 | 6.00 [4.16 to 8.66] | 1.43 [0.99 to 2.06] | 9.81 [5.29 to 18.19]
  6A | 13.86 [9.69 to 19.83] | 4.46 [2.18 to 9.12] | 7.37 [3.95 to 13.78]
  7F | 3.55 [2.35 to 5.36] | 1.23 [0.69 to 2.21] | 3.08 [1.72 to 5.51]
  19A | 13.07 [9.63 to 17.74] | 5.09 [3.17 to 8.19] | 10.50 [7.12 to 15.50]
Statistical Analysis 1: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; GMC ratio = 0.63, 95% CI 2-sided [0.23 to 1.76]
Statistical Analysis 2: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; GMC Ratio = 0.77, 95% CI 2-sided [0.30 to 1.99]
Statistical Analysis 3: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; GMC Ratio = 1.21, 95% CI 2-sided [0.38 to 3.86]
Statistical Analysis 4: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; [analysis description as in outcome 1, analysis 4]; Test type: Superiority or Other; GMC ratio = 0.93, 95% CI 2-sided [0.43 to 1.99]
Statistical Analysis 5: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 1, analysis 5]; Test type: Superiority or Other; GMC ratio = 1.09, 95% CI 2-sided [0.54 to 2.22]
Statistical Analysis 6: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 1, analysis 6]; Test type: Superiority or Other; GMC ratio = 1.18, 95% CI 2-sided [0.50 to 2.79]
Statistical Analysis 7: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; [analysis description as in outcome 1, analysis 7]; Test type: Superiority or Other; GMC ratio = 1.11, 95% CI 2-sided [0.56 to 2.19]
Statistical Analysis 8: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 1, analysis 8]; Test type: Superiority or Other; GMC ratio = 1.09, 95% CI 2-sided [0.58 to 2.06]
Statistical Analysis 9: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 1, analysis 9]; Test type: Superiority or Other; GMC ratio = 0.98, 95% CI 2-sided [0.46 to 2.13]
Statistical Analysis 10: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; [analysis description as in outcome 1, analysis 10]; Test type: Superiority or Other; GMC ratio = 0.98, 95% CI 2-sided [0.38 to 2.55]
Statistical Analysis 11: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 1, analysis 11]; Test type: Superiority or Other; GMC ratio = 1.23, 95% CI 2-sided [0.50 to 3.00]
Statistical Analysis 12: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 1, analysis 12]; Test type: Superiority or Other; GMC ratio = 1.25, 95% CI 2-sided [0.42 to 3.72]
Statistical Analysis 13: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; [analysis description as in outcome 1, analysis 13]; Test type: Superiority or Other; GMC ratio = 0.69, 95% CI 2-sided [0.29 to 1.68]
Statistical Analysis 14: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 1, analysis 14]; Test type: Superiority or Other; GMC ratio = 0.92, 95% CI 2-sided [0.40 to 2.10]
Statistical Analysis 15: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 1, analysis 15]; Test type: Superiority or Other; GMC ratio = 1.33, 95% CI 2-sided [0.49 to 3.64]
Statistical Analysis 16: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; [analysis description as in outcome 1, analysis 16]; Test type: Superiority or Other; GMC ratio = 1.70, 95% CI 2-sided [0.70 to 4.12]
Statistical Analysis 17: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 1, analysis 17]; Test type: Superiority or Other; GMC ratio = 1.37, 95% CI 2-sided [0.60 to 3.14]
Statistical Analysis 18: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 1, analysis 18]; Test type: Superiority or Other; GMC ratio = 0.81, 95% CI 2-sided [0.30 to 2.21]
Statistical Analysis 19: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; [analysis description as in outcome 1, analysis 19]; Test type: Superiority or Other; GMC ratio = 0.90, 95% CI 2-sided [0.43 to 1.89]
Statistical Analysis 20: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 1, analysis 20]; Test type: Superiority or Other; GMC ratio = 0.83, 95% CI 2-sided [0.42 to 1.67]
Statistical Analysis 21: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 1, analysis 21]; Test type: Superiority or Other; GMC ratio = 0.93, 95% CI 2-sided [0.40 to 2.16]
Statistical Analysis 22: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; [analysis description as in outcome 1, analysis 22]; Test type: Superiority or Other; GMC ratio = 7.53, 95% CI 2-sided [2.86 to 19.78]
Statistical Analysis 23: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 1, analysis 23]; Test type: Superiority or Other; GMC ratio = 0.53, 95% CI 2-sided [0.22 to 1.31]
Statistical Analysis 24: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 1, analysis 24]; Test type: Superiority or Other; GMC ratio = 0.07, 95% CI 2-sided [0.02 to 0.21]
Statistical Analysis 25: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; [analysis description as in outcome 1, analysis 25]; Test type: Superiority or Other; GMC ratio = 1.11, 95% CI 2-sided [0.53 to 2.30]
Statistical Analysis 26: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 1, analysis 26]; Test type: Superiority or Other; GMC ratio = 1.00, 95% CI 2-sided [0.50 to 1.97]
Statistical Analysis 27: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 1, analysis 27]; Test type: Superiority or Other; GMC ratio = 0.90, 95% CI 2-sided [0.39 to 2.07]
Statistical Analysis 28: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; [analysis description as in outcome 1, analysis 28]; Test type: Superiority or Other; GMC ratio = 4.20, 95% CI 2-sided [2.18 to 8.09]
Statistical Analysis 29: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 1, analysis 29]; Test type: Superiority or Other; GMC ratio = 0.61, 95% CI 2-sided [0.33 to 1.13]
Statistical Analysis 30: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 1, analysis 30]; Test type: Superiority or Other; GMC ratio = 0.15, 95% CI 2-sided [0.07 to 0.31]
Statistical Analysis 31: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; [analysis description as in outcome 1, analysis 31]; Test type: Superiority or Other; GMC ratio = 3.11, 95% CI 2-sided [1.51 to 6.40]
Statistical Analysis 32: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 1, analysis 32]; Test type: Superiority or Other; GMC ratio = 1.88, 95% CI 2-sided [0.96 to 3.69]
Statistical Analysis 33: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 1, analysis 33]; Test type: Superiority or Other; GMC ratio = 0.60, 95% CI 2-sided [0.27 to 1.37]
Statistical Analysis 34: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; [analysis description as in outcome 1, analysis 34]; Test type: Superiority or Other; GMC ratio = 2.88, 95% CI 2-sided [1.39 to 5.98]
Statistical Analysis 35: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 1, analysis 35]; Test type: Superiority or Other; GMC ratio = 1.15, 95% CI 2-sided [0.58 to 2.28]
Statistical Analysis 36: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 1, analysis 36]; Test type: Superiority or Other; GMC ratio = 0.40, 95% CI 2-sided [0.17 to 0.92]
Statistical Analysis 37: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; [analysis description as in outcome 1, analysis 37]; Test type: Superiority or Other; GMC ratio = 2.57, 95% CI 2-sided [1.50 to 4.39]
Statistical Analysis 38: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 1, analysis 38]; Test type: Superiority or Other; GMC ratio = 1.24, 95% CI 2-sided [0.75 to 2.05]
Statistical Analysis 39: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 1, analysis 39]; Test type: Superiority or Other; GMC ratio = 0.48, 95% CI 2-sided [0.26 to 0.89]

6. Secondary Outcome: Serotype-specific Opsonophagocytic Activity (OPA) Geometric Mean Titers (GMT) Prior to Single Dose of 13vPnC Vaccine
Description: Pneumococcal OPA GMTs for 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) were determined in the blood samples of all the participants using a microcolony OPA (mcOPA) assay. CIs for GMT are back transformations of a CI based on the Student t distribution for the mean logarithm of the titers.
Time Frame: Up to 7 days before vaccination
Population: Evaluable immunogenicity population. N= number of participants analyzed within a given treatment group. n= number of participants with a determinate OPA antibody titer to the given serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric mean titers
Arm/Group | 13vPnC/13vPnC/13vPnC | 7vPnC/7vPnC/13vPnC | 7vPnC/13vPnC/13vPnC
Number analyzed (Participants) | 44 | 18 | 22
Geometric mean titers
  4 (n= 40, 14, 19) | 8 [4.4 to 13.1] | 46 [7.8 to 268.5] | 45 [10.6 to 190.6]
  6B (n= 38, 16, 21) | 245 [92.6 to 646.9] | 247 [49.1 to 1241.8] | 332 [84.4 to 1304.3]
  9V (n= 40, 18, 21) | 43 [16.3 to 111.9] | 36 [8.6 to 149.1] | 52 [14.6 to 187.8]
  14 (n= 39, 16, 20) | 98 [39.7 to 242.9] | 40 [9.2 to 174.2] | 49 [14.4 to 163.9]
  18C (n= 42, 17, 19) | 14 [6.9 to 27.7] | 76 [15.7 to 363.0] | 28 [7.2 to 109.7]
  19F (n= 43, 17, 21) | 48 [20.8 to 112.5] | 49 [13.0 to 182.6] | 40 [14.0 to 112.5]
  23F (n= 43, 16, 21) | 52 [22.5 to 120.3] | 61 [13.1 to 284.3] | 178 [54.6 to 578.7]
  1 (n= 44, 18, 22) | 6 [4.5 to 7.5] | 5 [3.4 to 6.5] | 10 [6.9 to 15.0]
  3 (n= 42, 17, 21) | 20 [11.8 to 34.6] | 10 [4.4 to 22.2] | 18 [12.1 to 28.0]
  5 (n= 44, 18, 22) | 4 [NA to NA] — Since all values for serotype 5 in 13v/13v/13v treatment arm was less than lower limit of quantification (LLOQ), values was set to 0.5*limit of detection (LOD [8]) = 4. Hence variability (standard error) could not be estimated; CI was not estimable. | 4 [NA to NA] — Since all values for serotype 5 in 7v/7v/13v treatment arm was less than LLOQ, values was set to 0.5*LOD (8) = 4. Hence variability (standard error) could not be estimated; CI was not estimable. | 4 [3.6 to 5.6]
  6A (n= 44, 16, 21) | 170 [72.8 to 395.5] | 10 [3.4 to 31.4] | 75 [22.3 to 253.9]
  7F (n= 39, 16, 21) | 60 [22.5 to 157.8] | 47 [10.0 to 225.2] | 389 [112.0 to 1351.1]
  19A (n= 41, 18, 20) | 118 [58.2 to 239.7] | 25 [7.4 to 82.0] | 124 [46.4 to 330.2]
Statistical Analysis 1: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; Serotype 4: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/13vPnC/13vPnC - 7vPnC/7vPnC/13vPnC); Test type: Superiority or Other; GMT Ratio = 0.2, 95% CI 2-sided [0.04 to 0.73]
Statistical Analysis 2: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 4: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/13vPnC/13vPnC - 7vPnC/13vPnC/13vPnC); Test type: Superiority or Other; GMT Ratio = 0.2, 95% CI 2-sided [0.04 to 0.64]
Statistical Analysis 3: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 4: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (7vPnC/7vPnC/13vPnC - 7vPnC/13vPnC/13vPnC); Test type: Superiority or Other; GMT Ratio = 1.0, 95% CI 2-sided [0.19 to 5.46]
Statistical Analysis 4: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; Serotype 6B: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/13vPnC/13vPnC - 7vPnC/7vPnC/13vPnC); Test type: Superiority or Other; GMT ratio = 1.0, 95% CI 2-sided [0.17 to 5.85]
Statistical Analysis 5: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 6B: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/13vPnC/13vPnC - 7vPnC/13vPnC/13vPnC); Test type: Superiority or Other; GMT ratio = 0.7, 95% CI 2-sided [0.15 to 3.72]
Statistical Analysis 6: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 6B: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (7vPnC/7vPnC/13vPnC - 7vPnC/13vPnC/13vPnC); Test type: Superiority or Other; GMT ratio = 0.7, 95% CI 2-sided [0.10 to 5.37]
Statistical Analysis 7: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; Serotype 9V: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/13vPnC/13vPnC - 7vPnC/7vPnC/13vPnC); Test type: Superiority or Other; GMT ratio = 1.2, 95% CI 2-sided [0.23 to 6.25]
Statistical Analysis 8: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 9V: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/13vPnC/13vPnC - 7vPnC/13vPnC/13vPnC); Test type: Superiority or Other; GMT ratio = 0.8, 95% CI 2-sided [0.17 to 3.92]
Statistical Analysis 9: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 9V: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (7vPnC/7vPnC/13vPnC - 7vPnC/13vPnC/13vPnC); Test type: Superiority or Other; GMT ratio = 0.7, 95% CI 2-sided [0.11 to 4.43]
Statistical Analysis 10: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; Serotype 14: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/13vPnC/13vPnC - 7vPnC/7vPnC/13vPnC); Test type: Superiority or Other; GMT ratio = 2.4, 95% CI 2-sided [0.48 to 12.35]
Statistical Analysis 11: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 14: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/13vPnC/13vPnC - 7vPnC/13vPnC/13vPnC); Test type: Superiority or Other; GMT ratio = 2.0, 95% CI 2-sided [0.45 to 9.05]
Statistical Analysis 12: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 14: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (7vPnC/7vPnC/13vPnC - 7vPnC/13vPnC/13vPnC); Test type: Superiority or Other; GMT ratio = 0.8, 95% CI 2-sided [0.13 to 5.14]
Statistical Analysis 13: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; Serotype 18C: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/13vPnC/13vPnC - 7vPnC/7vPnC/13vPnC); Test type: Superiority or Other; GMT ratio = 0.2, 95% CI 2-sided [0.04 to 0.80]
Statistical Analysis 14: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 18C: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/13vPnC/13vPnC - 7vPnC/13vPnC/13vPnC); Test type: Superiority or Other; GMT ratio = 0.5, 95% CI 2-sided [0.12 to 2.03]
Statistical Analysis 15: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 18C: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (7vPnC/7vPnC/13vPnC - 7vPnC/13vPnC/13vPnC); Test type: Superiority or Other; GMT ratio = 2.7, 95% CI 2-sided [0.48 to 14.92]
Statistical Analysis 16: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; Serotype 19F: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/13vPnC/13vPnC - 7vPnC/7vPnC/13vPnC); Test type: Superiority or Other; GMT ratio = 1.0, 95% CI 2-sided [0.23 to 4.36]
Statistical Analysis 17: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 19F: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/13vPnC/13vPnC - 7vPnC/13vPnC/13vPnC); Test type: Superiority or Other; GMT ratio = 1.2, 95% CI 2-sided [0.31 to 4.84]
Statistical Analysis 18: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 19F: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (7vPnC/7vPnC/13vPnC - 7vPnC/13vPnC/13vPnC); Test type: Superiority or Other; GMT ratio = 1.2, 95% CI 2-sided [0.23 to 6.65]
Statistical Analysis 19: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; Serotype 23F: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/13vPnC/13vPnC - 7vPnC/7vPnC/13vPnC); Test type: Superiority or Other; GMT ratio = 0.9, 95% CI 2-sided [0.17 to 4.17]
Statistical Analysis 20: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 23F: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/13vPnC/13vPnC - 7vPnC/13vPnC/13vPnC); Test type: Superiority or Other; GMT ratio = 0.3, 95% CI 2-sided [0.07 to 1.24]
Statistical Analysis 21: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 23F: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (7vPnC/7vPnC/13vPnC - 7vPnC/13vPnC/13vPnC); Test type: Superiority or Other; GMT ratio = 0.3, 95% CI 2-sided [0.06 to 2.08]
Statistical Analysis 22: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; Serotype 1: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/13vPnC/13vPnC - 7vPnC/7vPnC/13vPnC); Test type: Superiority or Other; GMT ratio = 1.3, 95% CI 2-sided [0.79 to 1.97]
Statistical Analysis 23: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 1: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/13vPnC/13vPnC - 7vPnC/13vPnC/13vPnC); Test type: Superiority or Other; GMT ratio = 0.6, 95% CI 2-sided [0.38 to 0.88]
Statistical Analysis 24: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 1: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (7vPnC/7vPnC/13vPnC - 7vPnC/13vPnC/13vPnC); Test type: Superiority or Other; GMT ratio = 0.5, 95% CI 2-sided [0.27 to 0.77]
Statistical Analysis 25: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; Serotype 3: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/13vPnC/13vPnC - 7vPnC/7vPnC/13vPnC); Test type: Superiority or Other; GMT ratio = 2.0, 95% CI 2-sided [0.85 to 4.90]
Statistical Analysis 26: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 3: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/13vPnC/13vPnC - 7vPnC/13vPnC/13vPnC); Test type: Superiority or Other; GMT ratio = 1.1, 95% CI 2-sided [0.49 to 2.48]
Statistical Analysis 27: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 3: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (7vPnC/7vPnC/13vPnC - 7vPnC/13vPnC/13vPnC); Test type: Superiority or Other; GMT ratio = 0.5, 95% CI 2-sided [0.20 to 1.45]
Statistical Analysis 28: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; Serotype 5: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/13vPnC/13vPnC - 7vPnC/7vPnC/13vPnC); Test type: Superiority or Other; GMT ratio = 1.0, 95% CI 2-sided [0.87 to 1.15]
Statistical Analysis 29: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 5: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/13vPnC/13vPnC - 7vPnC/13vPnC/13vPnC); Test type: Superiority or Other; GMT ratio = 0.9, 95% CI 2-sided [0.79 to 1.03]
Statistical Analysis 30: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 5: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (7vPnC/7vPnC/13vPnC - 7vPnC/13vPnC/13vPnC); Test type: Superiority or Other; GMT ratio = 0.9, 95% CI 2-sided [0.76 to 1.06]
Statistical Analysis 31: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; Serotype 6A: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/13vPnC/13vPnC - 7vPnC/7vPnC/13vPnC); Test type: Superiority or Other; GMT ratio = 16.5, 95% CI 2-sided [3.56 to 76.14]
Statistical Analysis 32: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 6A: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/13vPnC/13vPnC - 7vPnC/13vPnC/13vPnC); Test type: Superiority or Other; GMT ratio = 2.3, 95% CI 2-sided [0.56 to 9.06]
Statistical Analysis 33: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 6A: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (7vPnC/7vPnC/13vPnC - 7vPnC/13vPnC/13vPnC); Test type: Superiority or Other; GMT ratio = 0.1, 95% CI 2-sided [0.02 to 0.78]
Statistical Analysis 34: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; Serotype 7F: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/13vPnC/13vPnC - 7vPnC/7vPnC/13vPnC); Test type: Superiority or Other; GMT ratio = 1.3, 95% CI 2-sided [0.22 to 7.07]
Statistical Analysis 35: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 7F: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/13vPnC/13vPnC - 7vPnC/13vPnC/13vPnC); Test type: Superiority or Other; GMT ratio = 0.2, 95% CI 2-sided [0.03 to 0.74]
Statistical Analysis 36: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 7F: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (7vPnC/7vPnC/13vPnC - 7vPnC/13vPnC/13vPnC); Test type: Superiority or Other; GMT ratio = 0.1, 95% CI 2-sided [0.02 to 0.84]
Statistical Analysis 37: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; Serotype 19A: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/13vPnC/13vPnC - 7vPnC/7vPnC/13vPnC); Test type: Superiority or Other; GMT ratio = 4.8, 95% CI 2-sided [1.35 to 16.98]
Statistical Analysis 38: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 19A: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/13vPnC/13vPnC - 7vPnC/13vPnC/13vPnC); Test type: Superiority or Other; GMT ratio = 1.0, 95% CI 2-sided [0.28 to 3.23]
Statistical Analysis 39: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 19A: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (7vPnC/7vPnC/13vPnC - 7vPnC/13vPnC/13vPnC); Test type: Superiority or Other; GMT ratio = 0.2, 95% CI 2-sided [0.05 to 0.85]

7. Secondary Outcome: Serotype-specific OPA GMTs 1 Month After Single Dose of 13vPnC Vaccine
Description: Serotype-specific pneumococcal OPA GMTs for the 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) were determined in the blood samples of all the participants using mcOPA assay. CIs for GMT are back transformations of a CI based on the Student t distribution for the mean logarithm of the titers.
Time Frame: One month after vaccination
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric mean titers
Arm/Group | 13vPnC/13vPnC/13vPnC | 7vPnC/7vPnC/13vPnC | 7vPnC/13vPnC/13vPnC
Number analyzed (Participants) | 120 | 57 | 58
Geometric mean titers
  4 (n= 117, 53, 55) | 5465 [4698.9 to 6356.4] | 5208 [4301.7 to 6304.2] | 5487 [4236.9 to 7106.4]
  6B (n= 117, 57, 56) | 6684 [5638.4 to 7924.4] | 10042 [7697.5 to 13101.6] | 8983 [7006.9 to 11516.8]
  9V (n= 116, 54, 55) | 5120 [4456.1 to 5882.6] | 4052 [3291.0 to 4989.7] | 5221 [4110.4 to 6630.7]
  14 (n= 115, 54, 55) | 2780 [2374.7 to 3254.6] | 3079 [2450.6 to 3869.4] | 2979 [2232.9 to 3973.4]
  18C (n= 117, 54, 57) | 7711 [6589.6 to 9023.3] | 7091 [5655.9 to 8889.9] | 8431 [6740.3 to 10545.7]
  19F (n= 118, 57, 57) | 1319 [1030.5 to 1689.5] | 1721 [1316.8 to 2250.3] | 1914 [1350.6 to 2712.5]
  23F (n= 118, 53, 56) | 2427 [2063.6 to 2855.0] | 2411 [1792.5 to 3242.4] | 2673 [2091.2 to 3417.3]
  1 (n= 119, 56, 57) | 613 [525.2 to 715.7] | 197 [161.4 to 239.4] | 1212 [968.0 to 1516.9]
  3 (n= 118, 56, 58) | 244 [214.7 to 276.4] | 173 [139.5 to 214.5] | 291 [239.4 to 353.7]
  5 (n= 118, 55, 54) | 455 [358.7 to 537.9] | 390 [281.2 to 541.8] | 728 [545.0 to 972.2]
  6A (n= 117, 55, 55) | 5580 [4593.6 to 6777.0] | 5596 [4276.6 to 7321.2] | 5982 [4450.7 to 8041.1]
  7F (n= 118, 56, 54) | 4323 [3794.4 to 4925.1] | 8048 [6500.9 to 9962.2] | 4056 [3092.2 to 5321.2]
  19A (n= 116, 53, 54) | 1212 [1048.1 to 1400.7] | 1249 [956.5 to 1632.3] | 1568 [1249.7 to 1966.1]
Statistical Analysis 1: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; GMT Ratio = 1.0, 95% CI 2-sided [0.80 to 1.38]
Statistical Analysis 2: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 6, analysis 2]; Test type: Superiority or Other; GMT Ratio = 1.0, 95% CI 2-sided [0.76 to 1.30]
Statistical Analysis 3: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 6, analysis 3]; Test type: Superiority or Other; GMT Ratio = 0.9, 95% CI 2-sided [0.69 to 1.30]
Statistical Analysis 4: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; [analysis description as in outcome 6, analysis 4]; Test type: Superiority or Other; GMT ratio = 0.7, 95% CI 2-sided [0.49 to 0.90]
Statistical Analysis 5: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 6, analysis 5]; Test type: Superiority or Other; GMT ratio = 0.7, 95% CI 2-sided [0.55 to 1.01]
Statistical Analysis 6: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 6, analysis 6]; Test type: Superiority or Other; GMT ratio = 1.1, 95% CI 2-sided [0.79 to 1.59]
Statistical Analysis 7: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; [analysis description as in outcome 6, analysis 7]; Test type: Superiority or Other; GMT ratio = 1.3, 95% CI 2-sided [0.98 to 1.63]
Statistical Analysis 8: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 6, analysis 8]; Test type: Superiority or Other; GMT ratio = 1.0, 95% CI 2-sided [0.76 to 1.27]
Statistical Analysis 9: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 6, analysis 9]; Test type: Superiority or Other; GMT ratio = 0.8, 95% CI 2-sided [0.58 to 1.05]
Statistical Analysis 10: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; GMT ratio = 0.9, 95% CI 2-sided [0.67 to 1.21]
Statistical Analysis 11: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 6, analysis 11]; Test type: Superiority or Other; GMT ratio = 0.9, 95% CI 2-sided [0.70 to 1.25]
Statistical Analysis 12: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 6, analysis 12]; Test type: Superiority or Other; GMT ratio = 1.0, 95% CI 2-sided [0.73 to 1.46]
Statistical Analysis 13: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; [analysis description as in outcome 6, analysis 13]; Test type: Superiority or Other; GMT ratio = 1.1, 95% CI 2-sided [0.83 to 1.43]
Statistical Analysis 14: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 6, analysis 14]; Test type: Superiority or Other; GMT ratio = 0.9, 95% CI 2-sided [0.70 to 1.20]
Statistical Analysis 15: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 6, analysis 15]; Test type: Superiority or Other; GMT ratio = 0.8, 95% CI 2-sided [0.61 to 1.15]
Statistical Analysis 16: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; [analysis description as in outcome 6, analysis 16]; Test type: Superiority or Other; GMT ratio = 0.8, 95% CI 2-sided [0.51 to 1.15]
Statistical Analysis 17: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 6, analysis 17]; Test type: Superiority or Other; GMT ratio = 0.7, 95% CI 2-sided [0.46 to 1.03]
Statistical Analysis 18: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 6, analysis 18]; Test type: Superiority or Other; GMT ratio = 0.9, 95% CI 2-sided [0.56 to 1.44]
Statistical Analysis 19: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; [analysis description as in outcome 6, analysis 19]; Test type: Superiority or Other; GMT ratio = 1.0, 95% CI 2-sided [0.74 to 1.37]
Statistical Analysis 20: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 6, analysis 20]; Test type: Superiority or Other; GMT ratio = 0.9, 95% CI 2-sided [0.67 to 1.23]
Statistical Analysis 21: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 6, analysis 21]; Test type: Superiority or Other; GMT ratio = 0.9, 95% CI 2-sided [0.63 to 1.29]
Statistical Analysis 22: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; [analysis description as in outcome 6, analysis 22]; Test type: Superiority or Other; GMT ratio = 3.1, 95% CI 2-sided [2.40 to 4.06]
Statistical Analysis 23: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 6, analysis 23]; Test type: Superiority or Other; GMT ratio = 0.5, 95% CI 2-sided [0.39 to 0.66]
Statistical Analysis 24: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 6, analysis 24]; Test type: Superiority or Other; GMT ratio = 0.2, 95% CI 2-sided [0.12 to 0.22]
Statistical Analysis 25: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; [analysis description as in outcome 6, analysis 25]; Test type: Superiority or Other; GMT ratio = 1.4, 95% CI 2-sided [1.11 to 1.78]
Statistical Analysis 26: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 6, analysis 26]; Test type: Superiority or Other; GMT ratio = 0.8, 95% CI 2-sided [0.66 to 1.06]
Statistical Analysis 27: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 6, analysis 27]; Test type: Superiority or Other; GMT ratio = 0.6, 95% CI 2-sided [0.45 to 0.78]
Statistical Analysis 28: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; [analysis description as in outcome 6, analysis 28]; Test type: Superiority or Other; GMT ratio = 1.2, 95% CI 2-sided [0.84 to 1.62]
Statistical Analysis 29: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 6, analysis 29]; Test type: Superiority or Other; GMT ratio = 0.6, 95% CI 2-sided [0.45 to 0.87]
Statistical Analysis 30: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 6, analysis 30]; Test type: Superiority or Other; GMT ratio = 0.5, 95% CI 2-sided [0.36 to 0.79]
Statistical Analysis 31: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; [analysis description as in outcome 6, analysis 31]; Test type: Superiority or Other; GMT ratio = 1.0, 95% CI 2-sided [0.71 to 1.40]
Statistical Analysis 32: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 6, analysis 32]; Test type: Superiority or Other; GMT ratio = 0.9, 95% CI 2-sided [0.66 to 1.31]
Statistical Analysis 33: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 6, analysis 33]; Test type: Superiority or Other; GMT ratio = 0.9, 95% CI 2-sided [0.63 to 1.39]
Statistical Analysis 34: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; [analysis description as in outcome 6, analysis 34]; Test type: Superiority or Other; GMT ratio = 0.5, 95% CI 2-sided [0.41 to 0.70]
Statistical Analysis 35: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 6, analysis 35]; Test type: Superiority or Other; GMT ratio = 1.1, 95% CI 2-sided [0.82 to 1.38]
Statistical Analysis 36: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 6, analysis 36]; Test type: Superiority or Other; GMT ratio = 2.0, 95% CI 2-sided [1.46 to 2.69]
Statistical Analysis 37: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; [analysis description as in outcome 6, analysis 37]; Test type: Superiority or Other; GMT ratio = 1.0, 95% CI 2-sided [0.74 to 1.28]
Statistical Analysis 38: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 6, analysis 38]; Test type: Superiority or Other; GMT ratio = 0.8, 95% CI 2-sided [0.59 to 1.02]
Statistical Analysis 39: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; [analysis description as in outcome 6, analysis 39]; Test type: Superiority or Other; GMT ratio = 0.8, 95% CI 2-sided [0.58 to 1.10]

8. Secondary Outcome: Percentage of Participants With at Least 1/8 Serotype-specific OPA GMTs After Single Dose of 13vPnC Vaccine
Description: Percentage of participants with at least 1/8 serotype-specific pneumococcal OPA GMTs for the 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) determined in the blood samples of all participants.
Time Frame: One month after vaccination
Population: The data was not collected as planned as the additional, more stringent qualification and validation of the improved mcOPA assays used in this study did not support 1/8 for the quantitation of a serum response and thus the established LLOQ was used for the mcOPA assay.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | 13vPnC/13vPnC/13vPnC | 7vPnC/7vPnC/13vPnC | 7vPnC/13vPnC/13vPnC
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Percentage of Participants With at Least 1/2048 OPA GMTs for Serotype 7F After Single Dose of 13vPnC Vaccine
Description: Percentage of participants with at least 1/2048 serotype-specific pneumococcal OPA GMTs for serotype 7F determined in the blood samples of all participants.
Time Frame: One month after vaccination
Population: The data was not collected as planned as the additional, more stringent qualification and validation of the improved mcOPA assays used in this study did not support 1/2048 for serotype 7F for the quantitation of a serum response and thus the established LLOQ was used for the mcOPA assay.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | 13vPnC/13vPnC/13vPnC | 7vPnC/7vPnC/13vPnC | 7vPnC/13vPnC/13vPnC
Number analyzed (Participants) | 0 | 0 | 0

10. Post Hoc Outcome: Percentage of Participants Achieving OPA GMTs With at Least Lower Limit of Quantification (LLOQ) 1 Month After Single Dose of 13vPnC Vaccine
Description: Percentage of participants achieving OPA GMTs with at least LLOQ for 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F and 23F) determined in blood samples of all participants using mcOPA assay. Exact 2-sided CI based on observed proportion of participants. LLOQ in titers for each serotype was: Pn001, 18; Pn003, 12; Pn004, 21; Pn005, 29; Pn06A, 37; Pn06B, 43; Pn7F, 210; Pn09V, 345; Pn014, 35; Pn18C, 31; Pn19A, 18; Pn19F, 48; Pn23F, 13. LOD established as lowest titer possible in assay, which was 8. OPA titers below LLOQ set to 0.5*LOD for analysis.
Time Frame: One month after vaccination
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | 13vPnC/13vPnC/13vPnC | 7vPnC/7vPnC/13vPnC | 7vPnC/13vPnC/13vPnC
Number analyzed (Participants) | 120 | 57 | 58
Percentage of Participants
  4 (n= 117, 53, 55) | 100.0 [96.9 to 100.0] | 100.0 [93.3 to 100.0] | 100.0 [93.5 to 100.0]
  6B (n= 117, 57, 56) | 100.0 [96.9 to 100.0] | 100.0 [93.7 to 100.0] | 100.0 [93.6 to 100.0]
  9V (n= 116, 54, 55) | 100.0 [96.9 to 100.0] | 100.0 [93.4 to 100.0] | 100.0 [93.5 to 100.0]
  14 (n= 115, 54, 55) | 100.0 [96.8 to 100.0] | 100.0 [93.4 to 100.0] | 100.0 [93.5 to 100.0]
  18C (n= 117, 54, 57) | 100.0 [96.9 to 100.0] | 100.0 [93.4 to 100.0] | 100.0 [93.7 to 100.0]
  19F (n= 118, 57, 57) | 98.3 [94.0 to 99.8] | 100.0 [93.7 to 100.0] | 98.2 [90.6 to 100.0]
  23F (n= 118, 53, 56) | 100.0 [96.9 to 100.0] | 100.0 [93.3 to 100.0] | 100.0 [93.6 to 100.0]
  1 (n= 119, 56, 57) | 100.0 [96.9 to 100.0] | 100.0 [93.6 to 100.0] | 100.0 [93.7 to 100.0]
  3 (n= 118, 56, 58) | 100.0 [96.9 to 100.0] | 98.2 [90.4 to 100.0] | 100.0 [93.8 to 100.0]
  5 (n= 118, 55, 54) | 99.2 [95.4 to 100.0] | 96.4 [87.5 to 99.6] | 100.0 [93.4 to 100.0]
  6A (n= 117, 55, 55) | 100.0 [96.9 to 100.0] | 100.0 [93.5 to 100.0] | 100.0 [93.5 to 100.0]
  7F (n= 118, 56, 54) | 100.0 [96.9 to 100.0] | 100.0 [93.6 to 100.0] | 100.0 [93.4 to 100.0]
  19A (n= 116, 53, 54) | 100.0 [96.9 to 100.0] | 100.0 [93.3 to 100.0] | 100.0 [93.4 to 100.0]
Statistical Analysis 1: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; Serotype 4: Difference in proportion, expressed as percentage, was calculated by percentage of participants achieving at least LLOQ in 13vPnC/13vPnC/13vPnC minus the percentage of participants achieving at least LLOQ in 7vPnC/7vPnC/13vPnC along with exact 2-sided 95% CI; Test type: Superiority or Other; Percent Difference = 0.0, 95% CI 2-sided [-3.5 to 6.7]
Statistical Analysis 2: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 4: Difference in proportion, expressed as percentage, was calculated by percentage of participants achieving at least LLOQ in 13vPnC/13vPnC/13vPnC minus the percentage of participants achieving at least LLOQ in 7vPnC/13vPnC/13vPnC along with exact 2-sided 95% CI; Test type: Superiority or Other; Percent Difference = 0.0, 95% CI 2-sided [-3.6 to 6.5]
Statistical Analysis 3: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 4: Difference in proportion, expressed as percentage, was calculated by percentage of participants achieving at least LLOQ in 7vPnC/7vPnC/13vPnC minus the percentage of participants achieving at least LLOQ in 7vPnC/13vPnC/13vPnC along with exact 2-sided 95% CI; Test type: Superiority or Other; Percent Difference = 0.0, 95% CI 2-sided [-6.8 to 6.6]
Statistical Analysis 4: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; Serotype 6B: Difference in proportion, expressed as percentage, was calculated by percentage of participants achieving at least LLOQ in 13vPnC/13vPnC/13vPnC minus the percentage of participants achieving at least LLOQ in 7vPnC/7vPnC/13vPnC along with exact 2-sided 95% CI; Test type: Superiority or Other; Percent Difference = 0.0, 95% CI 2-sided [-3.7 to 6.3]
Statistical Analysis 5: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 6B: Difference in proportion, expressed as percentage, was calculated by percentage of participants achieving at least LLOQ in 13vPnC/13vPnC/13vPnC minus the percentage of participants achieving at least LLOQ in 7vPnC/13vPnC/13vPnC along with exact 2-sided 95% CI; Test type: Superiority or Other; Percent difference = 0.0, 95% CI 2-sided [-3.6 to 6.4]
Statistical Analysis 6: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 6B: Difference in proportion, expressed as percentage, was calculated by percentage of participants achieving at least LLOQ in 7vPnC/7vPnC/13vPnC minus the percentage of participants achieving at least LLOQ in 7vPnC/13vPnC/13vPnC along with exact 2-sided 95% CI; Test type: Superiority or Other; Percent Difference = 0.0, 95% CI 2-sided [-6.4 to 6.5]
Statistical Analysis 7: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; Serotype 9V: Difference in proportion, expressed as percentage, was calculated by percentage of participants achieving at least LLOQ in 13vPnC/13vPnC/13vPnC minus the percentage of participants achieving at least LLOQ in 7vPnC/7vPnC/13vPnC along with exact 2-sided 95% CI; Test type: Superiority or Other; Percent Difference = 0.0, 95% CI 2-sided [-3.6 to 6.6]
Statistical Analysis 8: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 9V: Difference in proportion, expressed as percentage, was calculated by percentage of participants achieving at least LLOQ in 13vPnC/13vPnC/13vPnC minus the percentage of participants achieving at least LLOQ in 7vPnC/13vPnC/13vPnC along with exact 2-sided 95% CI; Test type: Superiority or Other; Percent Difference = 0.0, 95% CI 2-sided [-3.6 to 6.5]
Statistical Analysis 9: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 9V: Difference in proportion, expressed as percentage, was calculated by percentage of participants achieving at least LLOQ in 7vPnC/7vPnC/13vPnC minus the percentage of participants achieving at least LLOQ in 7vPnC/13vPnC/13vPnC along with exact 2-sided 95% CI; Test type: Superiority or Other; Percent Difference = 0.0, 95% CI 2-sided [-6.7 to 6.5]
Statistical Analysis 10: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; Serotype 14: Difference in proportion, expressed as percentage, was calculated by percentage of participants achieving at least LLOQ in 13vPnC/13vPnC/13vPnC minus the percentage of participants achieving at least LLOQ in 7vPnC/7vPnC/13vPnC along with exact 2-sided 95% CI; Test type: Superiority or Other; Percent Difference = 0.0, 95% CI 2-sided [-3.7 to 6.6]
Statistical Analysis 11: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 14: Difference in proportion, expressed as percentage, was calculated by percentage of participants achieving at least LLOQ in 13vPnC/13vPnC/13vPnC minus the percentage of participants achieving at least LLOQ in 7vPnC/13vPnC/13vPnC along with exact 2-sided 95% CI; Test type: Superiority or Other; Percent Difference = 0.0, 95% CI 2-sided [-3.7 to 6.5]
Statistical Analysis 12: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 14: Difference in proportion, expressed as percentage, was calculated by percentage of participants achieving at least LLOQ in 7vPnC/7vPnC/13vPnC minus the percentage of participants achieving at least LLOQ in 7vPnC/13vPnC/13vPnC along with exact 2-sided 95% CI; Test type: Superiority or Other; Percent Difference = 0.0, 95% CI 2-sided [-6.7 to 6.5]
Statistical Analysis 13: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; Serotype 18C: Difference in proportion, expressed as percentage, was calculated by percentage of participants achieving at least LLOQ in 13vPnC/13vPnC/13vPnC minus the percentage of participants achieving at least LLOQ in 7vPnC/7vPnC/13vPnC along with exact 2-sided 95% CI; Test type: Superiority or Other; Percent Difference = 0.0, 95% CI 2-sided [-3.6 to 6.6]
Statistical Analysis 14: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 18C: Difference in proportion, expressed as percentage, was calculated by percentage of participants achieving at least LLOQ in 13vPnC/13vPnC/13vPnC minus the percentage of participants achieving at least LLOQ in 7vPnC/13vPnC/13vPnC along with exact 2-sided 95% CI; Test type: Superiority or Other; Percent Difference = 0.0, 95% CI 2-sided [-3.7 to 6.3]
Statistical Analysis 15: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 18C: Difference in proportion, expressed as percentage, was calculated by percentage of participants achieving at least LLOQ in 7vPnC/7vPnC/13vPnC minus the percentage of participants achieving at least LLOQ in 7vPnC/13vPnC/13vPnC along with exact 2-sided 95% CI; Test type: Superiority or Other; Percent Difference = 0.0, 95% CI 2-sided [-6.6 to 6.4]
Statistical Analysis 16: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; Serotype 19F: Difference in proportion, expressed as percentage, was calculated by percentage of participants achieving at least LLOQ in 13vPnC/13vPnC/13vPnC minus the percentage of participants achieving at least LLOQ in 7vPnC/7vPnC/13vPnC along with exact 2-sided 95% CI; Test type: Superiority or Other; Percent Difference = -1.7, 95% CI 2-sided [-6.2 to 4.5]
Statistical Analysis 17: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 19F: Difference in proportion, expressed as percentage, was calculated by percentage of participants achieving at least LLOQ in 13vPnC/13vPnC/13vPnC minus the percentage of participants achieving at least LLOQ in 7vPnC/13vPnC/13vPnC along with exact 2-sided 95% CI; Test type: Superiority or Other; Percent Difference = 0.1, 95% CI 2-sided [-4.8 to 7.5]
Statistical Analysis 18: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 19F: Difference in proportion, expressed as percentage, was calculated by percentage of participants achieving at least LLOQ in 7vPnC/7vPnC/13vPnC minus the percentage of participants achieving at least LLOQ in 7vPnC/13vPnC/13vPnC along with exact 2-sided 95% CI; Test type: Superiority or Other; Percent Difference = 1.8, 95% CI 2-sided [-4.8 to 9.5]
Statistical Analysis 19: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; Serotype 23F: Difference in proportion, expressed as percentage, was calculated by percentage of participants achieving at least LLOQ in 13vPnC/13vPnC/13vPnC minus the percentage of participants achieving at least LLOQ in 7vPnC/7vPnC/13vPnC along with exact 2-sided 95% CI; Test type: Superiority or Other; Percent Difference = 0.0, 95% CI 2-sided [-3.5 to 6.7]
Statistical Analysis 20: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 23F: Difference in proportion, expressed as percentage, was calculated by percentage of participants achieving at least LLOQ in 13vPnC/13vPnC/13vPnC minus the percentage of participants achieving at least LLOQ in 7vPnC/13vPnC/13vPnC along with exact 2-sided 95% CI; Test type: Superiority or Other; Percent Difference = 0.0, 95% CI 2-sided [-3.6 to 6.4]
Statistical Analysis 21: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 23F: Difference in proportion, expressed as percentage, was calculated by percentage of participants achieving at least LLOQ in 7vPnC/7vPnC/13vPnC minus the percentage of participants achieving at least LLOQ in 7vPnC/13vPnC/13vPnC along with exact 2-sided 95% CI; Test type: Superiority or Other; Percent Difference = 0.0, 95% CI 2-sided [-6.7 to 6.5]
Statistical Analysis 22: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; Serotype 1: Difference in proportion, expressed as percentage, was calculated by percentage of participants achieving at least LLOQ in 13vPnC/13vPnC/13vPnC minus the percentage of participants achieving at least LLOQ in 7vPnC/7vPnC/13vPnC along with exact 2-sided 95% CI; Test type: Superiority or Other; Percent Difference = 0.0, 95% CI 2-sided [-3.5 to 6.4]
Statistical Analysis 23: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 1: Difference in proportion, expressed as percentage, was calculated by percentage of participants achieving at least LLOQ in 13vPnC/13vPnC/13vPnC minus the percentage of participants achieving at least LLOQ in 7vPnC/13vPnC/13vPnC along with exact 2-sided 95% CI; Test type: Superiority or Other; Percent Difference = 0.0, 95% CI 2-sided [-3.6 to 6.3]
Statistical Analysis 24: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 1: Difference in proportion, expressed as percentage, was calculated by percentage of participants achieving at least LLOQ in 7vPnC/7vPnC/13vPnC minus the percentage of participants achieving at least LLOQ in 7vPnC/13vPnC/13vPnC along with exact 2-sided 95% CI; Test type: Superiority or Other; Percent Difference = 0.0, 95% CI 2-sided [-6.5 to 6.3]
Statistical Analysis 25: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; Serotype 3: Difference in proportion, expressed as percentage, was calculated by percentage of participants achieving at least LLOQ in 13vPnC/13vPnC/13vPnC minus the percentage of participants achieving at least LLOQ in 7vPnC/7vPnC/13vPnC along with exact 2-sided 95% CI; Test type: Superiority or Other; Percent Difference = 1.8, 95% CI 2-sided [-1.7 to 9.6]
Statistical Analysis 26: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 3: Difference in proportion, expressed as percentage, was calculated by percentage of participants achieving at least LLOQ in 13vPnC/13vPnC/13vPnC minus the percentage of participants achieving at least LLOQ in 7vPnC/13vPnC/13vPnC along with exact 2-sided 95% CI; Test type: Superiority or Other; Percent Difference = 0.0, 95% CI 2-sided [-3.7 to 6.2]
Statistical Analysis 27: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 3: Difference in proportion, expressed as percentage, was calculated by percentage of participants achieving at least LLOQ in 7vPnC/7vPnC/13vPnC minus the percentage of participants achieving at least LLOQ in 7vPnC/13vPnC/13vPnC along with exact 2-sided 95% CI; Test type: Superiority or Other; Percent Difference = -1.8, 95% CI 2-sided [-9.6 to 4.5]
Statistical Analysis 28: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; Serotype 5: Difference in proportion, expressed as percentage, was calculated by percentage of participants achieving at least LLOQ in 13vPnC/13vPnC/13vPnC minus the percentage of participants achieving at least LLOQ in 7vPnC/7vPnC/13vPnC along with exact 2-sided 95% CI; Test type: Superiority or Other; Percent Difference = 2.8, 95% CI 2-sided [-2.0 to 11.3]
Statistical Analysis 29: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 5: Difference in proportion, expressed as percentage, was calculated by percentage of participants achieving at least LLOQ in 13vPnC/13vPnC/13vPnC minus the percentage of participants achieving at least LLOQ in 7vPnC/13vPnC/13vPnC along with exact 2-sided 95% CI; Test type: Superiority or Other; Percent Difference = -0.8, 95% CI 2-sided [-4.9 to 5.6]
Statistical Analysis 30: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 5: Difference in proportion, expressed as percentage, was calculated by percentage of participants achieving at least LLOQ in 7vPnC/7vPnC/13vPnC minus the percentage of participants achieving at least LLOQ in 7vPnC/13vPnC/13vPnC along with exact 2-sided 95% CI; Test type: Superiority or Other; Percent Difference = -3.6, 95% CI 2-sided [-12.5 to 3.2]
Statistical Analysis 31: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; Serotype 6A: Difference in proportion, expressed as percentage, was calculated by percentage of participants achieving at least LLOQ in 13vPnC/13vPnC/13vPnC minus the percentage of participants achieving at least LLOQ in 7vPnC/7vPnC/13vPnC along with exact 2-sided 95% CI; Test type: Superiority or Other; Percent Difference = 0.0, 95% CI 2-sided [-3.6 to 6.5]
Statistical Analysis 32: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 6A: Difference in proportion, expressed as percentage, was calculated by percentage of participants achieving at least LLOQ in 13vPnC/13vPnC/13vPnC minus the percentage of participants achieving at least LLOQ in 7vPnC/13vPnC/13vPnC along with exact 2-sided 95% CI; Test type: Superiority or Other; Percent Difference = 0.0, 95% CI 2-sided [-3.6 to 6.5]
Statistical Analysis 33: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 6A: Difference in proportion, expressed as percentage, was calculated by percentage of participants achieving at least LLOQ in 7vPnC/7vPnC/13vPnC minus the percentage of participants achieving at least LLOQ in 7vPnC/13vPnC/13vPnC along with exact 2-sided 95% CI; Test type: Superiority or Other; Percent Difference = 0.0, 95% CI 2-sided [-6.6 to 6.6]
Statistical Analysis 34: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; Serotype 7F: Difference in proportion, expressed as percentage, was calculated by percentage of participants achieving at least LLOQ in 13vPnC/13vPnC/13vPnC minus the percentage of participants achieving at least LLOQ in 7vPnC/7vPnC/13vPnC along with exact 2-sided 95% CI; Test type: Superiority or Other; Percent Difference = 0.0, 95% CI 2-sided [-3.6 to 6.4]
Statistical Analysis 35: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 7F: Difference in proportion, expressed as percentage, was calculated by percentage of participants achieving at least LLOQ in 13vPnC/13vPnC/13vPnC minus the percentage of participants achieving at least LLOQ in 7vPnC/13vPnC/13vPnC along with exact 2-sided 95% CI; Test type: Superiority or Other; Percent Difference = 0.0, 95% CI 2-sided [-3.5 to 6.6]
Statistical Analysis 36: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 7F:Difference in proportion, expressed as percentage, was calculated by percentage of participants achieving at least LLOQ in 7vPnC/7vPnC/13vPnC minus the percentage of participants achieving at least LLOQ in 7vPnC/13vPnC/13vPnC along with exact 2-sided 95% CI; Test type: Superiority or Other; Percent Difference = 0.0, 95% CI 2-sided [-6.5 to 6.7]
Statistical Analysis 37: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/7vPnC/13vPnC; Serotype 19A: Difference in proportion, expressed as percentage, was calculated by percentage of participants achieving at least LLOQ in 13vPnC/13vPnC/13vPnC minus the percentage of participants achieving at least LLOQ in 7vPnC/7vPnC/13vPnC along with exact 2-sided 95% CI; Test type: Superiority or Other; Percent Difference = 0.0, 95% CI 2-sided [-3.6 to 6.7]
Statistical Analysis 38: Comparison: 13vPnC/13vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 19A: Difference in proportion, expressed as percentage, was calculated by percentage of participants achieving at least LLOQ in 13vPnC/13vPnC/13vPnC minus the percentage of participants achieving at least LLOQ in 7vPnC/13vPnC/13vPnC along with exact 2-sided 95% CI; Test type: Superiority or Other; Percent Difference = 0.0, 95% CI 2-sided [-3.6 to 6.6]
Statistical Analysis 39: Comparison: 7vPnC/7vPnC/13vPnC vs 7vPnC/13vPnC/13vPnC; Serotype 19A: Difference in proportion, expressed as percentage, was calculated by percentage of participants achieving at least LLOQ in 7vPnC/7vPnC/13vPnC minus the percentage of participants achieving at least LLOQ in 7vPnC/13vPnC/13vPnC along with exact 2-sided 95% CI; Test type: Superiority or Other; Percent Difference = 0.0, 95% CI 2-sided [-6.8 to 6.6]

ADVERSE EVENTS:
Time Frame: AEs/SAEs: recorded from signing of informed consent form to completion of study (28-42 days post 13vPnC). Participants recorded prespecified AEs in electronic diary:local reactions; systemic events; use of antipyretic medication (Day 1-Day 7 post 13vPnC).
Description: SAEs and AEs were grouped by system organ class and summarized. AEs included solicited AEs collected in the electronic diary (local and systemic reactions; systematic assessment) and unsolicited events collected on the case report form at each visit (nonsystematic assessment).
Arm/Group | 13vPnC/13vPnC/13vPnC | 7vPnC/7vPnC/13vPnC | 7vPnC/13vPnC/13vPnC
Serious Adverse Events (participants affected / at risk) | 0/130 | 0/64 | 0/64
Other Adverse Events (participants affected / at risk) | 82/130 | 36/64 | 39/64
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | 13vPnC/13vPnC/13vPnC (N=130) | 7vPnC/7vPnC/13vPnC (N=64) | 7vPnC/13vPnC/13vPnC (N=64)
Pain (Any) (Skin and subcutaneous tissue disorders) | 62/112 | 29/52 | 34/53 — Pain (Any) = present at site of vaccination
Pain (Mild) (Skin and subcutaneous tissue disorders) | 55/109 | 25/51 | 29/51 — Pain (Mild) = does not interfere with activity
Pain (Moderate) (Skin and subcutaneous tissue disorders) | 17/95 | 12/47 | 10/48 — Pain (Moderate) = interferes with activity
Pain (Severe) (Skin and subcutaneous tissue disorders) | 1/90 | 1/43 | 1/45 — Pain (Severe) = prevents daily activity
Swelling (Any) (Skin and subcutaneous tissue disorders) | 40/101 | 20/48 | 13/47 — Swelling (Any) = present at site of vaccination
Swelling (Mild) (Skin and subcutaneous tissue disorders) | 27/96 | 17/48 | 11/47 — Swelling (Mild) = 0.5 - 2.0 cm
Swelling (Moderate) (Skin and subcutaneous tissue disorders) | 24/97 | 9/44 | 5/46 — Swelling (Moderate) = 2.5 - 7.0 cm
Swelling (Severe) (Skin and subcutaneous tissue disorders) | 0/90 | 1/43 | 0/45 — Swelling (Severe) = >7.0 cm
Redness (Any) (Skin and subcutaneous tissue disorders) | 51/105 | 27/50 | 23/50 — Redness (Any) = present at site of vaccination
Redness (Mild) (Skin and subcutaneous tissue disorders) | 39/101 | 20/49 | 18/48 — Redness (Mild) = 0.5 - 2.0 cm
Redness (Moderate) (Skin and subcutaneous tissue disorders) | 21/95 | 14/45 | 8/47 — Redness (Moderate) = 2.5 - 7.0 cm
Redness (Severe) (Skin and subcutaneous tissue disorders) | 0/90 | 1/43 | 0/45 — Redness (Severe) = >7.0 cm
Fever >= 38.0 degree C but <=39.0 degree C (General disorders) | 14/93 | 14/49 | 9/46
Fever >39.0 to <=40.0 degree C (General disorders) | 2/92 | 2/43 | 1/46
Fever >40.0 degree C (General disorders) | 0/90 | 0/43 | 1/45
Vomiting (Any) (General disorders) | 3/91 | 4/44 | 3/45 — Vomiting (Any) = present
Vomiting (Mild) (General disorders) | 3/91 | 4/44 | 3/45 — Vomiting (Mild)= 1-2 times in 24 hours
Vomiting (Moderate) (General disorders) | 0/90 | 0/43 | 0/45 — Vomiting (Moderate) = >2 times in 24 hours
Vomiting (Severe) (General disorders) | 0/90 | 0/43 | 0/45 — Vomiting (Severe) = requires IV hydration
Diarrhea (Any) (General disorders) | 8/90 | 8/45 | 4/47 — Diarrhea (Any) = present
Diarrhea (Mild) (General disorders) | 8/90 | 8/45 | 4/47 — Diarrhea (Mild) = 2-3 loose stools in 24 hours
Diarrhea (Moderate) (General disorders) | 1/90 | 0/43 | 0/45 — Diarrhea (Moderate) = 4-5 stools in 24 hours
Diarrhea (Severe) (General disorders) | 0/90 | 0/43 | 0/45 — Diarrhea (Severe) = 6 or more loose stools in 24 hours
Fatigue (Any) (General disorders) | 42/103 | 28/54 | 15/48 — Fatigue (Any) = present
Fatigue (Mild) (General disorders) | 34/100 | 17/49 | 10/48 — Fatigue (Mild) = does not interfere with activity
Fatigue (Moderate) (General disorders) | 16/96 | 15/49 | 7/46 — Fatigue (Moderate) = some interference with activity
Fatigue (Severe) (General disorders) | 3/92 | 1/43 | 1/45 — Fatigue (Severe) = prevents daily routine activity
Injection site erythema (General disorders) | 1 | 0 | 0
Acute tonsillitis (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 2 | 0 | 0
Ear infection (Infections and infestations) | 0 | 1 | 1
Gastroenteritis (Infections and infestations) | 1 | 1 | 1
Nasopharyngitis (Infections and infestations) | 3 | 0 | 0
Pharyngitis (Infections and infestations) | 2 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 2 | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Varicella (Infections and infestations) | 2 | 0 | 1
Viral infection (Infections and infestations) | 2 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.